

# **Clinical Trial Protocol**

Doc. No.: c02543230-04 1315.1 **BI Trial No.: BI Investigational** BI 836858 **Product:** A Phase I, open-label, cohort dose escalation trial with BI 836858 in patients Title: with refractory or relapsed acute myeloid leukemia and patients with acute myeloid leukemia in complete remission with high risk to relapse **Clinical Phase:** I **Trial Clinical** Monitor: Phone: Fax: **Co-ordinating Investigator:** Phone: Fax: Revised Protocol (based on Global Amendments 01, 02, and 03) **Status: Version and Date:** Version: 4.0 **Date: 28 APRIL 2016**  Proprietary confidential information.

 $\hbox{@ 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies. All rights reserved.}$ 

This document may not - in full or in part - be passed on, reproduced, published or otherwise used without prior written permission.

## CLINICAL TRIAL PROTOCOL SYNOPSIS

| Name of company: | | | Tabulated | |
|---|---|---|---|---|
| Boehringer Ingelheim | | | Trial Protocol | |
| Name of finished produ | ct: | | | |
| Not applicable | | | | |
| Name of active ingredie | ent: | | | |
| BI 836858 | | | | |
| Protocol date: | Trial r | umber: | | Revision date: |
| 21 DEC 2011 | 1315.1 | | | 28 APRIL 2016 |
| Title of trial: | refracto | ry or relapsed ac | ohort dose escalation trial with BI 83<br>ute myeloid leukemia and patients v<br>mission with high risk to relapse | |
| Co-ordinating | | | | |
| Investigator: | | | | |
| | 25.11 | | | |
| Trial sites: | Multi-centre trial | | | |
| Clinical phase: | I | | | |
| Objectives: | To investigate the maximum tolerated dose (MTD), safety and tolerability, pharmacokinetics and efficacy of BI 836858 monotherapy in acute myeloid leukemis (AML) patients with refractory or relapsed AML and patients with AML in complet remission (CR) with high risk to relapse | | | |
| Methodology: | | bel cohort dose | | |
| No. of patients: | Planned | number: about 6 | 53 | |
| total entered: | About 3 | 6 (for refractory | or relapsed AML) and 27 (for AML | patients in CR) |
| each treatment: | About 3 | -6 (per dose cohe | ort, for each patient population) | |
| Diagnosis : | Acute N | Iyeloid Leukemi | a | |
| Main criteria | Adult p | atients with relap | osed or refractory AML | |
| for inclusion: | AND | | | |
| | Patients | with AML in CI | R with high risk to relapse defined a | s: |
| | a) | LeukemiaNet (I<br>induction and callogeneic hema<br>available, not el | with non-favorable genetics (according ELN) classification) that are in CR at consolidation chemotherapy and are atopoietic stem cell transplantation (ligible/fit enough) | after having received not candidates for |
| | <b>b</b> ) | Of AMI patients u | with non-favorable genetics (according | ng to ELN classification) |
| | b) | | vith non-favorable genetics (according allogeneic hematopoietic stem | |


28 Apr 2016

| Doc. No.: c02543230-04 | Trial Protocol |
|------------------------|----------------|

| Name of company: | | Tabulated<br>Trial Protocol | |
|---|---|---|---|
| Boehringer Ingelheim | | | |
| Name of finished produ | ict: | | |
| Not applicable | | | |
| Name of active ingredie | ent: | | |
| BI 836858 | | | |
| Protocol date: | Trial number: | | Revision date: |
| 21 DEC 2011 | 1315.1 | | 28 APRIL 2016 |
| Test product: | BI 836858 | | |
| dose: | The starting dose for BI | 836858 will be | |
| | - 10 mg for refrac | ctory or relapsed AML patients and | |
| | _ | patients in CR with high risk to rel | apse |
| mode of admin.: | Intravenous (i.v.) infusio | on | |
| Comparator products: | Not applicable | | |
| Duration of treatment: | Patients with refractory | or relapsed AML | |
| | | up to 8 repeated administrations as le | ong as neither patient nor |
| | Investigator requests trea | | Vanlain a Crasson (IWC) as |
| | | nefit, defined by the International Wese (partial remission (PR) or comple | |
| | complete remission with | incomplete blood recovery (CRi)) of | or subjective response (in |
| | | response) after 8 administrations an until progressive disease (PD) | d who are tolerating the |
| | infusions, may continue | uniti progressive disease (FD) | |
| | AML patients in CR with | h high risk to relapse | |
| | The first three administra | ations will be given every second w | eek, on day 1 of Cycles 1, |
| | 2 and 3. From the 4 <sup>th</sup> ad | ministration onwards, patients will i | receive monthly (every |
| | | of BI 836858 (i.e. 4 <sup>th</sup> infusion on Cy<br>for overall up to one year of treatmen | |
| | relapse or infusions are r | | nt unitess these patients |
| | | repeated administrations as long as r | neither patient nor |
| C * | Investigator requests trea | | |
| Criteria for efficacy: | | l, time to treatment failure<br>coverall response | |
| | | 1 | to refractory or relapsed |
| | AML patients. AML patients in CR. | | applies only to |
| Criteria for safety: | * | e, incidence and intensity of adverse | events graded according |
| Cintila idi Salety. | | ogy criteria for adverse events (CTC | - |
| | incidence of dose-limiting | ng toxicity, vital signs, ECG, physica | |
| G4-4*-4*1 41 1 | laboratory parameters. | | |
| Statistical methods: | Descriptive statistics. | | |


# FLOW CHART - A (REFRACTORY OR RELAPSED PATIENTS)

| Trial Periods | Screen | Treatment* | | | | EOT | Furth | FU | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | Screen | (1 | Cycle 1<br>Cycle | – Cycl<br>= 14 da | e 4<br>ays) | ЕОТ | F | ГЕ | EOFT | FU |
| Visit | 1 | Cx<br>V1 | Cx<br>V2 | Cx<br>V3 | Cx<br>V4 | | Cx<br>V1 | Cx<br>V2 | | |
| Days<br>(in respective cycle)* | -14 to - | 1 | 4<br>±1 <sup>1</sup> | 8 | 11<br>±1 <sup>1</sup> | | 1 | 8 | | |
| Informed consent | Х | | | | | | | | | |
| Informed consent for pharmacogenetics | Х | | | | | | | | | |
| Demographics and baseline conditions | Х | | | | | | | | | |
| Medical history | Х | | | | | | | | | |
| Review of in-/exclusion criteria | х | x <sup>2</sup> | | | | | | | | |
| Dose assignment | x 3 | | | | | | | | | |
| LABS/SAFETY ASSESSMI | | | | | | | <u> </u> | | : | |
| Safety laboratory parameters incl. urinalysis <sup>4</sup> | Х | X | x <sup>1</sup> | X | x <sup>1</sup> | Х | Х | Х | X | X |
| Physical examination<br>ECOG performance status | X | x <sup>5</sup> | | | | Х | x <sup>5</sup> | | х | X |
| Vital signs, height <sup>6</sup> , weight <sup>6</sup> | X | X | Х | X | Х | X | X | X | X | X |
| Serum pregnancy test <sup>7</sup> | X | X | | | | X | X | | X | |
| 12 lead-ECG | X | X | | | | X | | | x <sup>8</sup> | |
| Adverse events | X | X | X | X | X | X | X | X | X | X |
| Concomitant therapy DISEASE ASSESSMENTS | X | X | X | X | X | X | Х | X | X | x <sup>9</sup> |
| Bone marrow aspiration | X | x <sup>10</sup> | | $\mathbf{x}^{10}$ | | x <sup>11</sup> | | | x <sup>8, 11</sup> | x 11 |
| -<br>- | | | | | | | <u> </u> | | | |
| _ | | | <u> </u> | | <u> </u> | <u> </u> | <u> </u> | | <u> </u> | |
| <u> </u> | <u> </u> | | L _ | | <u> </u> | <u> </u> | <u> </u> | | <u> </u> | |
| _ | <u> </u> | | ┞ │ | | | <u> </u> | <u> </u> | | <u> </u> | |
| TRIAL MEDICATION | | | | | | | | | | |
| Drug Administration | | X | | X | | | Х | Х | | |
| Eligibility for further administration | | x <sup>16</sup> | | x <sup>16</sup> | | x <sup>16,17</sup> | X <sup>16, 17</sup> | x <sup>16, 17</sup> | | |
| End of active trial treatment | | | | | | X | | | | |
| End of further treatment | | | | | | | | | X | |
| Other therapy for AML | | | | | | | | | | X |
| Vital Status | | | | | | | | | | X |

Boehringer Ingelheim 28 Apr 2016 BI Trial No.: 1315.1

- EOT: End of treatment evaluation, including an evaluation for further treatment. Those patients with clinical benefit, PR, CRi, or CR after 8 administrations and who are tolerating the infusions well may continue until PD or other criteria for withdrawal are met as noted in Section 3.3.4.1. For those patients who will receive more than 8 administrations, this visit is to be performed 7 days (±2 days) after the 8<sup>th</sup> administration of BI 836858. For those patients who receive ≤ 8 administrations, this visit is to be performed 14 days (±2 days) after the last administration of BI 836858.
- FTE: Further treatment evaluation. Each patient who will receive more than 8 administrations will have a FTE visit for each infusion. The visit numbers are 6, 7, 8, etc. until the patient discontinues.
- EOFT: End of further treatment. For each patient who receives more than 8 administrations, there will be an end of further treatment evaluation. This visit is to be performed 14 days (±2 days) after the last administration of BI 836858.
- FU: Follow-up, starts after the last administration of BI 836858, visits at least every 4 weeks until 6 months after the last administration of BI 836858.
- \* The planned duration of a treatment cycle is 14 days; there will be two administrations of BI 836858 per cycle.
- \*\* These visits are only for those patients with clinical benefit, PR, CRi or CR after 8 administrations and who are tolerating the infusions well who continue until PD or other criteria for withdrawal are met as noted in Section 3.3.4.1.
- 1 Visit window of ±1 day only allowed beginning in Cycle 3 and for all subsequent cycles. In Cycles 1 and 2 visit window not allowed due to the PK schedule as outlined in <u>Tables 1a</u> and <u>2a</u>.
- 2 Review of inclusion/exclusion criteria during screening and again on day of first administration.
- 3 After informed consent and review of inclusion/exclusion criteria (timing described in footnote 2).
- For details refer to Section 5.2.3.1. Urine has to be measured only at screening, EOT, EOFT and FU visits. Safety laboratory assessments may be completed up to 2 days prior to administration. An additional safety lab will be collected on day 2 (i.e., 24 hours after the first administration of BI 836858). Other lab tests to be included: Haptoglobin, direct antiglobulin test, bilirubin (direct and indirect) and free hemoglobin.
- Only every second cycle (i.e. before cycle 1, 3, 5, 7 etc.) Physical examination may be completed up to 2 days prior to administration. Eastern Cooperative Oncology Group (ECOG) score must be completed on the day of the administration. If the first administration of BI 836858 occurs within 3 days of the screening visit, these examinations do not need to be repeated.
- 6 Height and weight only at day 1 of first administration of BI 836858; weight also at EOT and EOFT.
- For women of childbearing potential only. Serum pregnancy test is to be completed at odd numbered administrations only (e.g. administration 1, 3, 5, etc.).
- 8 ECG, bone marrow aspiration, tests will be performed at EOFT only if the patient has completed at least 2 cycles (e.g. received 4 administrations) since the EOT visit.
- 9 Concomitant therapy during FU is collected only if indicated for treatment of adverse event.
- Bone marrow aspirate to assess efficacy before 5<sup>th</sup> and 9<sup>th</sup> administrations (i.e., BM performed on Day 1 (+/- 1) of cycles 3 and 5 and treatment started on day 1 (up to +3 days) of cycles 3 and 5) (see Section 5.1.2).
- Only one sample to be collected at the time of PD or the time of initiation of other anti-leukemia therapy, which may be at the EOT/EOFT, if PD or initiation of other anti-leukemia therapy occurs during treatment, or during follow-up. If the patient is non-progressing/not receiving other anti-leukemia therapy at the end of follow-up or the trial, the sample will be obtained at the last follow-up visit for this patient.

- 16 Can be performed up to 2 days prior to this visit.
- After the 8<sup>th</sup> infusion, at the end of treatment visit, patients will be evaluated to determine if they have clinical benefit, as defined by IWG objective response (PR, CRi or CR) or subjective response (in the absence of objective response) and are tolerating the infusions well and who would like to continue to receive infusions until PD or other criteria for withdrawal are met as noted in Section 3.3.4.1. For each infusion past the 8<sup>th</sup> administration, patients will continue to be assessed after each cycle for clinical benefit (objective or subjective response), and that they are tolerating the infusions well and would like to continue until PD or other criteria for withdrawal are met as noted in Section 3.3.4.1.


# FLOW CHART - B (AML PATIENTS IN CR)

| Trial Periods | Screen | Tr | eatmer | ıt* | | Further<br>tment* | | End of<br>Treatment | End of Residual<br>Effect Period<br>and Follow-up 1 | Follow-up |
|---|---|---|---|---|---|---|---|---|---|---|
| | | Cycle 1 – Cycle 3<br>(1 Cycle = 14 days) | | FTE<br>(every 2nd cycle;<br>Cycles 5, 7, 921) | | ЕоТ | EoR/FU1 | FU2 to FU6 | | |
| Visit | 1 | Cx<br>V1 | Cx<br>V2 | Cx<br>V3 | Cx<br>V1 | Cx<br>V2 | Cx<br>V3 | As soon as possible<br>but not later than<br>one week after<br>permanent<br>discontinuation of<br>trial medication | Not earlier than 30<br>days after permanent<br>discontinuation of<br>trial medication | Every 4<br>weeks |
| Days (in respective cycle)*1 | -14 to<br>-1 | 1 | 2 | 8 | 1 | 2 | 8 | | | |
| Informed consent | Х | | | | | | | | | |
| Informed consent for pharmacogenetics | Х | | | | | | | : | : | :<br> |
| Demographics and baseline conditions | Х | | | | | | | | | |
| Medical history | Х | | | | | | | | | |
| Review of incl-/excl criteria | х | x <sup>2</sup> | | | | | | <u> </u> | <u> </u> | |
| Dose assignment | x <sup>3</sup> | | | | | | | | | |
| LABS/SAFETY<br>ASSESSMENTS | | | | | | | | <u> </u> | <u> </u> | |
| Safety laboratory parameters incl. urinalysis <sup>4</sup> | х | Х | Х | | Х | | | х | Х | х |
| Physical examination and ECOG performance status <sup>5</sup> | Х | x <sup>5</sup> | :<br>:<br>:<br>:<br>:<br>:<br>:<br>: | | x <sup>5</sup> | | | х | | х |
| Vital signs, height <sup>6</sup> , weight <sup>6</sup> | Х | X | х | | X | | | Х | X | X |
| Serum pregnancy test <sup>7</sup> | Х | X | | | Х | | | Х | | |
| 12 lead-ECG | Х | X | | | X | | | Х | x <sup>8</sup> | |
| Adverse events | Х | X | Х | Х | Х | Х | х | Х | Х | Х |
| Concomitant therapy | х | х | Х | Х | Х | х | х | х | х | x <sup>9</sup> |
| DISEASE ASSESSMENT | | | | | | | | | | |
| Bone marrow (BM) aspiration 10 | X | х | | | | | | x | | Х |
| _ | | | | | | | | | | |
| Disease assessment w/ PB and clinical assessment | | Х | | | Х | | | х | | |
| Disease assessment w/ BM or biopsy 12 | | x | | | Х | | | x | | |
| · | • | <u> </u> | <u> </u> | <u> </u> | <del></del> | | $\vdash$ $-$ | | | |
| <del>.</del> ——— | | $\vdash$ | <u> </u> | | | | | <u> </u> | | |
| | $\vdash \vdash$ | $\vdash$ | | | <b>—</b> — | | | | | |
| TRIAL MEDICATION | | | | | | | | | | |
| Drug Administration | | Х | | | Х | | | X | | |
| Eligibility for further administration | | Х | | | x <sup>16</sup> | | | | | |
| End of active trial treatment | | | | | | | | Х | | |
| Other therapy for AML | | | <del></del> | | | | | X | X | Х |
| Vital Status | | | | | | | | | | Х |


© 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies. All rights reserved.

This document may not - in full or in part - be passed on, reproduced, published or otherwise used without prior written permission.

Boehringer Ingelheim BI Trial No.: 1315.1 Doc. No.: c02543230-04 28 Apr 2016


EOT: End of treatment evaluation. The EOT visit will be performed as soon as possible but no later than one week (7

days) after permanent discontinuation of trial medication for any reason, or when the Investigator decides with the

Trial Protocol

patient to permanently discontinue the trial medication.

FTE: Further treatment evaluation. Each patient who will receive more than 3 administrations will have a FTE visit for each infusion. The visits are completed on day 1 of every second cycle (i.e. 5, 7, 9, etc.) until the patient discontinues or completes up to 12 months of therapy. Infusions are every 2 weeks for the first 3 cycles then for FTE, these treatments are monthly.

EoR: The End of Residual End Period visit should not be performed earlier than 30 days after permanent discontinuation of the trial medication.

- FU: Follow-up visits after the last administration of BI 836858 completed, at least every 4 weeks until 6 months after the last administration of BI 836858. In case patients do not visit the site, the FU visit can be conducted by phone.
- \* The planned duration of a treatment cycle is 14 days; there will be one administration of BI 836858
- \*\* These visits are only for those patients after 3 administrations and who are tolerating the infusions well who continue until PD or other criteria for withdrawal are met as noted in <u>Section 3.3.4.1</u>. These visits occur every second cycle (i.e., Cycles 5, 7, 9...21)
- Visit window of  $\pm 1$  day only allowed beginning in Cycle 9. In Cycles 1 through 7 visit window not allowed due to the PK schedule as outlined in <u>Tables 1b</u> and <u>2b</u>.
- 2 Review of inclusion/exclusion criteria during screening and again on day of first administration.
- 3 After informed consent and review of inclusion/exclusion criteria (timing described in footnote 2).
- For details refer to Section 5.2.3.1. Urine has to be measured only at screening, FTE, EOT and FU visits. Safety laboratory assessments may be completed up to 2 days prior to administration. An additional safety lab will be collected on day 2 (i.e., 24 hours after the first administration of BI 836858). Other lab tests to be included: Haptoglobin, direct antiglobulin test, bilirubin (direct and indirect) and free hemoglobin.
- At screening and every second cycle (i.e. before cycle 1, 3, 5, 7 etc.) Physical examination may be completed up to 2 days prior to administration. Eastern Cooperative Oncology Group (ECOG) score must be completed on the day of the administration. If the first administration of BI 836858 occurs within 3 days of the screening visit, these examinations do not need to be repeated.
- 6 Height and weight only at day 1 of first administration of BI 836858; weight also at EOT.
- For women of childbearing potential only. Serum pregnancy test to be completed at odd numbered administrations only (e.g., administration 1, 3, 5, etc.)
- 8 ECG will be performed at visit 1 of each cycle and at EoR if abnormal at EOT.
- 9 Concomitant therapy during FU is collected only if indicated for treatment of adverse event.
- Bone marrow aspirate to be performed, at investigator discretion, if there is suspicion of relapse.
- Disease assessment with bone marrow (or biopsy) is to be performed if suspicion of relapse
- 16 Can be performed up to 2 days prior to this visit.

28 Apr 2016

| | | _ | | | Т | <br>_ | | _ |
|---|---|---|---|---|---|---|---|---|
| _ | <br> | | | | L | <br> | _ | |
| | | | - | | Γ ' | | | |
| | | _ | | - | † | <br> | <u> </u> | |
| | | _ | | | - | | _ | |
| | | _ | | | ┡ . | <br> | | |
| | | _ | _ | | L | <br>_ | | |
| | | | _ | | L | <br><u>_</u> | | |
| | <br> | - | - | | T | _ | | |
| | | _ | | | + . | | <del> </del> | |
| | | _ | | - | <b>├</b> . | <br><del>-</del> - | <u> </u> | |








Doc. No.: c02543230-04 Trial Protocol 





## **TABLE OF CONTENTS**

| TTI | | 'AGE | I |
|---|---|---|---|
| CL | INIC | AL TRIAL PROTOCOL SYNOPSIS | 2 |
| | ow ( | CHART - A (REFRACTORY OR RELAPSED | |
| | | TIENTS) | |
| | | CHART - B (AML PATIENTS IN CR) | |
| TA | BLE | OF CONTENTS | . 13 |
| AB | BRE | VIATIONS | . 18 |
| 1. | INT | RODUCTION | . 22 |
| | 1.1 | MEDICAL BACKGROUND | |
| | 1.2 | DRUG PROFILE | |
| 2. | RA | ΓΙΟΝΑLE, OBJECTIVES, AND BENEFIT - RISK | |
| | | ESSMENT | . 26 |
| | 2.1 | RATIONALE FOR PERFORMING THE TRIAL | |
| | 2.2 | TRIAL OBJECTIVES | |
| | 2.3 | BENEFIT - RISK ASSESSMENT | 27 |
| 3. | DES | SCRIPTION OF DESIGN AND TRIAL POPULATION | . 30 |
| | 3.1 | OVERALL TRIAL DESIGN AND PLAN | 30 |
| | | 3.1.1 Administrative structure of the trial | 31 |
| | 3.2 | DISCUSSION OF TRIAL DESIGN, INCLUDING THE CHOICE OF CONTROL GROUP | |
| | 3.3 | SELECTION OF TRIAL POPULATION | |
| | | 3.3.1 Main diagnosis for study entry | 33 |
| | | 3.3.2 Inclusion criteria | |
| | | 3.3.3 Exclusion criteria | |
| | | 3.3.4 Removal of patients from therapy or assessments | |
| | | 3.3.4.1 Removal of individual patients | |
| 4. | TRI | EATMENTS | |
| ٠. | 4.1 | TREATMENTS TO BE ADMINISTERED | |
| | 4.1 | 4.1.1 Identity of BI investigational product and comparator product | |
| | | 4.1.2 Method of assigning patients to treatment groups | |
| | | 4.1.3 Selection of doses in the trial | |
| | | 4.1.4 Drug assignment and administration of doses for each patient | |


| | | 4.1.5 | Blinding and procedures for unblinding | 43 |
|---|---|---|---|---|
| | | | 4.1.5.1 Blinding | 43 |
| | | | 4.1.5.2 Procedures for emergency unblinding | 43 |
| | | 4.1.6 | Packaging, labelling, and re-supply | 43 |
| | | 4.1.7 | Storage conditions | 43 |
| | | 4.1.8 | Drug accountability | 44 |
| | 4.2 | | COMITANT THERAPY, RESTRICTIONS, AND RESCUE | 44 |
| | | 4.2.1 | Rescue medication, emergency procedures, and additional treatments | 44 |
| | | 4.2.2 | Restrictions | |
| | | | 4.2.2.1 Restrictions regarding concomitant treatment | |
| | | | 4.2.2.2 Restrictions on diet and life style | |
| | 4.3 | TREA | ATMENT COMPLIANCE | |
| <b>5.</b> | | | ES AND THEIR ASSESSMENT | |
| J. | | | | |
| | 5.1 | | CACY – PHARMACODYNAMICS | |
| | | 5.1.1 | Endpoints of efficacy | |
| | | 5.1.2 | Assessment of efficacy | ,4 / |
| | | | 5.1.2.3 Assessment and definition of best overall response | 48 |
| | | | 5.1.2.4 Progression free survival (PFS) | 49 |
| | | | 5.1.2.5 Time to treatment failure (TTF) | 50 |
| | 5.2 | | TY | |
| | | 5.2.1 | Endpoints of safety | |
| | | | 5.2.1.1 Dose limiting toxicity (DLT) for refractory or relapse patients | 51 |
| | | | 5.2.1.2 Dose limiting toxicity (DLT) for AML patients in CR | 52 |
| | | 5.2.2 | Assessment of adverse events | 53 |
| | | | 5.2.2.1 Definitions of AEs | 53 |
| | | | 5.2.2.2 Adverse event collection and reporting | 56 |
| | | 5.2.3 | Assessment of safety laboratory parameters | 58 |
| | | | 5.2.3.1 General safety laboratory parameters | 58 |
| | | 5.2.4 | Electrocardiogram | |
| | | 5.2.5 | Assessment of other safety parameters | 60 |


| | 5.2.5.1 | Vital signs | 60 |
|------------|-------------------|-----------------------|----|
| | 5.2.5.2 | Physical examination | 60 |
| <b>5.4</b> | <b>APPROPRIAT</b> | ENESS OF MEASUREMENTS | 60 |

| <b>6.</b> | INV | ESTIC | GATION | NAL PLAN | 66 |
|---|---|---|---|---|---|
| | 6.1 | VISIT | SCHED | ULE | 66 |
| | <b>6.2</b> | .2 DETAILS OF TRIAL PROCEDURES AT SELECTED VISITS | | | |
| | | <b>6.2.1</b> | Screeni | ng and run-in period | 66 |
| | | <b>6.2.2</b> | Treatm | ent periods for refractory or relapsed AML patients | 67 |
| | | | 6.2.2.1 | Visit 1 and Visit 3 – day of BI 836858 administration (administrations 1-8) | 67 |
| | | | 6.2.2.2 | Visit 2 and Visit 4 (+ 1 day window allowed beginning in Cycle 3), following administration of BI 836858 | 68 |
| | 6.2.3 End of treatment and follow-up period for refractory or | | | | |
| | | | relapse | d AML patients | 68 |
| | | | 6.2.3.1 | EOT visit | 68 |
| | | | 6.2.3.2 | Further treatment (Visit 1 and Visit 2) | 69 |
| | | | 6.2.3.3 | End of further treatment | 70 |
| | | 6.2.4 | Treatm | ent period for AML patients in CR | 70 |
| | | | 6.2.4.1 | Visit 1– Day 1 of BI 836858 administration (administration 3) | |
| | | | 6.2.4.2 | Further treatment. | |
| | | | 6.2.4.3 | End of Treatment (EOT) visit | 72 |


BI Trial No.: 1315.1 Doc. No.: c02543230-04

| | | 6.2.4.4 End of Residual Effect Period visit (EoR) | 72 |
|---|---|---|---|
| | | 6.2.5 Follow up | |
| | | 6.2.6 End of the whole trial | 73 |
| <b>7.</b> | | ATISTICAL METHODS AND DETERMINATION OF MPLE SIZE | 75 |
| | 7.1 | STATISTICAL DESIGN - MODEL | |
| | 7.1 | NULL AND ALTERNATIVE HYPOTHESES | |
| | | PLANNED ANALYSES | |
| | 7.3 | 7.3.1 Primary analyses | |
| | | 7.3.2 Secondary analyses | |
| | | 7.5.2 Secondary analyses | |
| | | 7.3.2.3 Best overall response | 76 |
| | | 7.3.2.4 Progression free survival, time to treatment failure, | |
| | | 7.3.3 Safety analyses | 77 |
| | | 7.3.4 Interim analyses | 77 |
| | 7.4 | HANDLING OF MISSING DATA | |
| | 7.5 | RANDOMISATION | |
| | <b>7.6</b> | DETERMINATION OF SAMPLE SIZE | 80 |
| 8. | | ORMED CONSENT, DATA PROTECTION, TRIAL | |
| | RE | CORDS | 81 |
| | 8.1 | STUDY APPROVAL, PATIENT INFORMATION, AND INFORME CONSENT | |
| | 8.2 | DATA QUALITY ASSURANCE | 81 |
| | 8.3 | RECORDS | |
| | | 8.3.1 Source documents | 82 |
| | | 8.3.2 Direct access to source data and documents | |
| | 8.4 | LISTEDNESS AND EXPEDITED REPORTING OF ADVERSE | |
| | | EVENTS | 83 |
| | | 8.4.1 Listedness | |
| | | 8.4.2 Expedited reporting to health authorities and IECs/IRBs | 83 |


Boehringer Ingelheim 28 Apr 2016 BI Trial No.: 1315.1

| JI 111a1 110 1515.1 | |
|------------------------|----------------|
| Doc. No : c02543230-04 | Trial Protocol |

| | 8.5 | STATEMENT OF CONFIDENTIALITY | 83 |
|---|---|---|---|
| 9. | REFERENCES | | |
| | 9.1 | PUBLISHED REFERENCES | 84 |
| | 9.2 | UNPUBLISHED REFERENCES | 87 |
| 10. | APPENDICES | | |
| | 10.1 | PUBLICATION POLICIES | 88 |
| | 10.2 | EASTERN COOPERATIVE ONCOLOGY GROUP (ECOG) PERFORMANCE STATUS | 88 |
| | 10.3 | CLINICAL EVALUATION OF LIVER DISEASE | 89 |
| | | 10.3.1 Introduction | 89 |
| | | 10.3.2 Procedures | 89 |
| 11. | DES | CRIPTION OF GLOBAL AMENDMENTS | 91 |

## **ABBREVIATIONS**

AE Adverse Event

AESI Adverse event of special interest

ALT Alanine amino transferase

AML Acute myeloid leukemia

AMP Auxiliary medicinal product

ANC Absolute neutrophil count

anti-HB Hepatitis B surface antibody

anti-HCV Hepatitis C antibody AP Alkaline phosphatase

APL Acute promyelocytic leukemia

aPTT Activated partial thromboplastin time

AST Aspartate amino transferase

ASCT Allogeneic stem cell transplantation

BI Boehringer Ingelheim

BLO Below the lower limit of quantification

BM Bone marrow

CA Competent Authority

∘C Degree Celcius

CL Total plasma clearance

C<sub>max</sub> Maximum measured plasma concentration

CML Local Clinical Monitor
CNS Central nervous system
CR Complete Remission


CRi Complete Remission with incomplete blood recovery

CRA Clinical Research Associate

CRF Case Report Form

CRO Clinical Research Organization

CTCAE Common Terminology Criteria for Adverse Events

CTMF Clinical Trial Master File
CTP Clinical Trial Protocol
CTR Clinical Trial Report

DEDP Drug exposure during pregnancy

DILI Drug Induced Liver Injury
DLT Dose Limiting Toxicity
DNA Deoxyribonucleic-acid

eCRF Electronic Case Report Form

ECG Electrocardiogram

ECOG Eastern Cooperative Oncology Group

EDTA Ethylen-diamine-tetraacetic acid

ELN European LeukemiaNet
EOFT End of further treatment

EoR End of Residual Effect Period

EOT End of active treatment

FDA Food and Drug Administration
FTE Further treatment evaluation

FU Follow-up

GCP Good Clinical Practice

G-CSF Granulocyte colony stimulating factor

GvHD Graft versus Host Disease
HBsAg Hepatitis B surface antigen

HIV Human immunodeficiency virus


28 Apr 2016

IB Investigator's Brochure

ICH International Conference on Harmonization

IEC Independent Ethics Committee

INR International normalized ratio
IRB Institutional Review Board
IRR Infusion-related reaction
ISF Investigator Site File

i.v. Intravenous

IWG International Working Group

LDH Lactate dehydrogenase LFT Liver function test

mAB Monoclonal antibody

mg milligram

MTD Maximum Tolerated Dose

MedDRA Medical Dictionary for Drug Regulatory Activities

MRT Mean residence time
NBE New biological entity

NC Not calculated

NIMP Non-investigational medicinal product

NK Natural killer (cells)

NOA Not analyzed

NOP No peak detectable

NOR No valid result

NOS No sample available

OPU Operative Unit

ORR Objective Response Rate

PD Progressive disease

PFS Progression free survival

PK Pharmacokinetics

PLT Platelets

PR Partial Remission
PT Prothrombin time

REP Residual Effect Period; after the last dose of medication with measureable

drug levels or pharmacodynamic effects still likely to be present

RNA Ribonucleic-acid

RTPCR Reverse transcription polymerase chain reaction

SAE Serious Adverse Event

sCD33 Soluble CD33

SCT Stem cell transplantation

SD Stable disease

SDV Source data verification

SOP Standard Operating Procedure

SUSAR Suspected unexpected serious adverse reaction

TCM Trial Clinical Monitor

TDMAP Trial Data Management and Analysis Plan

TF Treatment Failure

TNF Tissue necrosis factor
TTF Time to treatment failure
ULN Upper limit of normal

WBC White blood cell count

WHO World Health Organization

Doc. No.: c02543230-04 Trial Protocol 

#### 1. INTRODUCTION

#### 1.1 MEDICAL BACKGROUND

Acute myeloid leukemia (AML) is a heterogeneous clonal disorder of hematopoietic progenitor cells and represents the most common malignant myeloid disorder in adults, with a prevalence of 3.8 cases per 100,000 rising to 17.9 cases per 100,000 adults aged 65 years and older (R07-2768). The median age at presentation is about 70 years, and three men are affected for every two women. Without therapeutic intervention the disease progresses and leads to death within months after initial diagnosis (R07-2768).

Genetic alterations in leukemic cells constitute the most important factor for the prognosis of AML (R07-2768, R07-2770, R07-2774). AML patients are classified in groups of favorable, intermediate, and unfavorable risk. Other factors with impact on prognosis are age, performance score, white blood cell count, blood chemistry disturbances and de-novo versus secondary AML.

Intensive treatment approaches for AML with curative intention include two phases. The first, induction treatment, most commonly consists of cytarabine and an anthracycline, is aiming to reach a CR. The second phase, post-remission treatment, is aiming to consolidate remission. AML patients under the age of 60 years achieve complete remission rates of up to 75 % following intensive treatment regimens, while AML patients over 60 years of age (referred to as elderly patients) have a 40 - 60 % chance of CR when receiving intensive remission induction treatment (R07-2767).

While the majority of younger AML patients receive intensive treatment, a substantial number of elderly patients are considered ineligible for this treatment approach (R07-2773, R07-2854). Therefore, the CR rates up to 60 % reported in elderly previously untreated AML patients receiving intensive treatment are by no means representative of the entire group of elderly AML patients. For AML patients considered ineligible to receive intensive treatment investigational treatments is widely regarded as the preferred therapeutic option (R07-2769, R07-2772). With these non-approved drugs CR rates up to 20 % are observed in randomized Phase III trials. Although patients who are considered as ineligible for intensive treatment constitute a generally accepted subgroup of AML patients, no validated criteria are defined to judge a patient's eligibility for intensive treatment (R07-2771). The assessment of eligibility for intensive treatment is performed regularly for every single patient based on the specialised physician's clinical experience and the comprehensive review of factors such as patient age, performance score, organ dysfunctions and co-morbidities, as well as the patient's informed decision.

The median overall survival (OS), for patients not achieving a CR is <1 year, even with best palliative treatment. Even for patients who have received induction and consolidation treatment the OS and cure rate are poor: Over 60 % will die due to their disease within 5 years. The risk of leukemic relapse along with the poor prospects of long-term survival after a relapse calls for novel therapeutic strategies to maintain CR in AML.

Boehringer Ingelheim BI Trial No.: 1315.1 Doc. No.: c02543230-04 28 Apr 2016


AML patients in CR who have been initially diagnosed with non-favorable genetics and either have received induction and consolidation treatment and are not candidates for allogeneic hematopoietic stem cell transplantation (e.g. no donor available, not eligible/fit enough) or have received an allogeneic hematopoietic stem cell transplantation have a very high risk to relapse. For those patients no standard therapy to maintain the CR is currently available.

**Trial Protocol** 

For refractory or relapsed AML patients, outside of treatment in clinical trials, re-induction followed by allogeneic stem cell transplantation is the most common regimen. However many are not eligible for such an intensive treatment. For those patients with refractory or relapsed AML ineligible for intensive treatment, or for those with refractory or relapses disease after allogeneic stem cell transplantation, no approved or standard treatment is available.

Evidence that targeting of CD33 can result in clinical benefit for patients suffering from AML is provided by the unconjugated, humanized IgG1 monoclonal antibody lintuzumab (SGN-33, HuM195) which showed signs of clinical efficacy as monotherapy in a Phase I clinical trial in relapsed / refractory AML patients with an objective response rate (ORR) of 17 % (R11-1481). Objective response was defined as either CR, CRi or PR.

Lintuzumab was also explored in a Phase I study in patients with acute promyelocytic leukemia (APL) after remission induction. Multiple doses of lintuzumab could be administered safely and appeared to eliminate minimal residual disease detectable by RTPCR in some patients. (R11-4695)

Currently, major efforts are focused on the improvement of the therapy in these subgroups of patients with unfavourable prognosis.

#### 1.2 DRUG PROFILE

BI 836858 is a fully human IgG1 antibody specific for human CD33 which is Fc-engineered for increased binding to FcγRIIIa. Please see full details in latest version of Investigator's Brochure (c02324887-03).

CD33 is a myeloid differentiation antigen which is expressed on the cell surface of non-malignant leukocytes of the myeloid lineage and with high frequency on malignant cells in AML, chronic myeloid leukemia and myelodysplastic syndrome (R11-1467, R11-1468, R11-1470, R11-2960). In addition to expression on malignant myeloid blast cells, CD33 expression was reported for leukemic stem cells (R11-1469). For normal leukocytes, CD33 expression was reported for monocytes, macrophages, dendritic cells, and to a lower extent, granulocytes (R11-1467), but not for CD34<sup>+</sup>CD38<sup>-</sup> hematopoietic stem cells in the bone marrow (R11-1469). Based on the expression profile of CD33, transient pharmacodynamic effects of CD33 antibody treatment on CD33 positive normal cell types may be expected.

Boehringer Ingelheim BI Trial No.: 1315.1 Doc. No.: c02543230-04 28 Apr 2016

Trial Protocol 

BI 836858 is Fc-engineered for increased binding to Fc $\gamma$ RIIIa, which results in increased antibody dependent cellular cytotoxicity (ADCC) activity of BI 836858 as compared to a non-Fc-engineered IgG1-type of antibody. The ADCC activity of BI 836858 was assessed on a panel of AML-derived cell lines and primary AML cells and compared to the ADCC activity of lintuzumab, a humanized CD33-specific antibody which has been in clinical development for AML (R11-1471).

The CD33 antigen is known to internalize upon antibody binding (R11-4256).

Preliminary data from this first-in-human dose escalation study with BI 836858 (trial number 1315.1) in patients with relapsed or refractory acute myeloid leukemia investigating a weekly dose (q1w) is available. As of the data cut-off date 12 April 2016, 26 patients were treated with BI 836858, all with doses of 10, 20 and 40 mg, respectively. The most frequent drug-related AE Preferred Term (PT) was infusion-related reaction (IRR) in eleven out of 26 patients (42 %). Adverse events considered a sign or symptom of an IRR by the investigator included back pain, chest pain, chills, dyspnea, fever and hypotension. All patients recovered from their IRRs with adequate symptom-oriented therapy. Drug-related transient increase of liver function tests was reported in four patients: one patient with grade 1 aspartate amino


Boehringer Ingelheim
28 Apr 2016
BI Trial No.: 1315.1

transferase (AST) and alanine amino transferase (ALT), one patient with grade 1 ALT, grade 3 AST and grade 3 bilirubin, one patient with grade 3 AST, grade 3 ALT and no increase of bilirubin and another one (not yet entered in the database) with grade 3 AST, grade 1 ALT and no increase of bilirubin.

Trial Protocol 

# 2. RATIONALE, OBJECTIVES, AND BENEFIT - RISK ASSESSMENT

#### 2.1 RATIONALE FOR PERFORMING THE TRIAL

New therapeutic strategies are needed to significantly improve the prognosis of AML patients with relapsed/refractory disease, but also for AML patients in CR with a high risk to relapse. Recent successful developments of signal transduction inhibitors or antibodies targeting specific molecules that are deemed important for the malignant cell biology have spurred the search for other targets and respective antibodies.

CD33 is a valid target to treat patients with AML, as CD33 is expressed on the majority of AML cells (R11-1472) and on leukemic stem cells, but not outside of the hematopoietic system (R11-1473).

CD 33 targeting approaches have been evaluated in clinical trials in AML patients. Gemtuzumab Ozogamicin (Mylotarg®), an immunoconjugate of a CD 33 mAb and calicheamicin, was approved by the Food and Drug Administration (FDA) in 2000 for patients over the age of 60 with relapsed AML, or those who are not considered candidates for standard chemotherapy. In June 2010 Mylotarg® was withdrawn by FDA request, due to a negative benefit risk assessment in a Phase III trial. As Mylotarg is an immunconjugate of a CD 33 mAb and a toxin, the MoA and also the safety profile are different to BI 836858. Clinical data of relapsed/refractory AML patients who were treated with the humanized CD33 IgG1 monoclonal antibody (mAb) lintuzumab are published (R11-1474, R01-1267, R11-1481). In these trials, administration of lintuzumab was safe and has shown signs of clinical efficacy (ORR) of 17 % in a Phase I trial in relapsed / refractory AML (R11-1481). Lintuzumab was also explored in a Phase I study in patients with APL after remission induction. Multiple doses of lintuzumab could be administered safely and appeared to eliminate minimal residual disease detectable by RTPCR in some patients. (R11-4695)

The clinical experience with lintuzumab supports the assumption that targeting CD33 with an IgG1-type antibody may translate into clinical benefit in patients with AML with an acceptable side effect profile.

BI 836858 is a monoclonal antibody which mechanistically relies on effector-cell mediated immune mechanisms, in particular ADCC (antibody dependent cellular cytotoxicity) and ADCP (antibody dependent cellular phagocytosis). ADCC predominantly depends on the presence of natural killer (NK) cells and ADCP on the presence of myeloid derived effector cells (i.e. monocytes and macrophages). In a recent publication, where NK cell phenotype and function was assessed in 32 consecutive AML patients including 12 achieving complete remission, it was reported that NK cells in relapsed and refractory AML patients have impaired functionality. It was also shown that phenotypic and functional abnormalities of NK cells are partially restored in AML patients achieving a CR. (R15-6192).

28 Apr 2016

It is likely that BI 836858 requires the presence of functional NK cells and monocytes to achieve clinical benefit in AML patients. AML patients who have achieved a CR have an improved effector cell profile (NK cells and monocytes) and may have a higher likelihood to benefit from the pharmacological activity of BI 836858.

This trial was the first administration of BI 836858 in humans.

#### 2.2 TRIAL OBJECTIVES

The primary objective of this trial is to determine the maximum tolerated doses (MTDs) of BI 836858. BI 836858 is a new biological entity (NBE) and the MTD may not be reached. To learn more about the safety and preliminary efficacy there will be an expansion cohort either at the MTD or the highest tested dose (e.g. 320 mg). Secondary objectives are to document the safety and tolerability of BI 836858,

and to evaluate efficacy (see Section 5).

## 2.3 BENEFIT - RISK ASSESSMENT

Although considerable progress has been achieved in understanding the etiology and biologic behavior of AML and the development of more effective treatment regimens are ongoing,


most patients with refractory or relapsed AML have a very poor prognosis. Re-induction followed by allogeneic stem cell transplantation is the most common regimen for refractory or relapsed AML patients, however many are not eligible for such an intensive treatment. For those patients with refractory or relapsed AML ineligible for intensive treatment, or for those with refractory or relapsed disease after allogeneic stem cell transplantation, no approved or standard treatment is available.

AML patients in CR who have been initially diagnosed with non-favorable genetics and either have received induction and consolidation treatment and are not candidates for allogeneic hematopoietic stem cell transplantation (e.g. no donor available, not eligible/fit enough) or have received an allogeneic hematopoietic stem cell transplantation have a very high risk to relapse. For those patients no standard therapy to maintain the CR is currently available.

BI 836858 is a monoclonal antibody, which specifically targets CD33. Targeting CD33 in patients with AML may potentially offer a benefit to those patients since CD33 is expressed on AML blasts in the majority of AML patients (see <a href="Section 1.2">Section 1.2</a>). *In vitro*, BI 836858 is a potent inducer of ADCC, which results in cytolysis of AML-derived cell lines and primary AML blasts from peripheral blood and bone marrow. In the clinical setting, these effects may potentially result in anti-leukemic activity as a monotherapy, but also offer potential for combination with other drugs in patients with AML.

CD33 is not known to be expressed outside of the hematopoietic system. The anticipated side effect profile of BI 836858 based on the CD33 expression profile comprises predominantly hematologic adverse events such as neutropenia. These hematological adverse events are frequently reported in patients with hematological diseases and may be due to the underlying disease, the treatment or both. The preclinical safety assessments for BI 836858 have revealed TNF-alpha and INF-gamma release, suggesting a potential for infusion reactions.

Clinical data from 26 patients are available from this first in human study 1315.1.

Infusion reactions were the most frequently observed drug related adverse event in this first in human study and is newly classified as a listed (expected) adverse event. Infusion-related reactions are frequently observed with monoclonal antibodies in hematological indications, and signs/symptoms of IRRs reported for BI 836858 are in line with AEs reported for other antibodies approved in hematology indications. To mitigate the risk for IRRs, protocol specified precautions must be adhered to, i.e. premedication, rate-controlled infusion schedule and symptom monitoring. If an IRR occurs the infusion of BI 836858 should be paused and additional supportive measures are recommended based on standard of care, e.g. additional corticosteroid or non-steroidal analgesics and/or opioids.in. So far no case of life-threatening IRR was reported; however in case a patient is developing a life-threatening IRR despite appropriate premedication the patient should discontinue the treatment with BI 836858 permanently. Drug-related transient increase of LFT was reported in 4 patients. In none of these cases Hy's law criteria were met. Frequent testing of LFTs is mandated during treatment with BI 836858 (frequency defined in the clinical trial protocols). In case of

Boehringer Ingelheim 28 Apr 2016 BI Trial No.: 1315.1

alterations of liver laboratory parameters the clinical evaluation of liver disease and follow up on liver laboratory parameters should be done as outlined in the clinical trial protocol.

Patients with refractory or relapsed AML with limited or no standard treatment options may benefit from blast cell reduction and disease stabilization following treatment with BI 836858. AML patients in CR who have been initially diagnosed with non-favorable genetics with a very high risk to relapse with limited or no standard treatment options may benefit from targeting CD33 positive leukemic stem cells and maintenance of achieved complete remission to initial standard therapy.

The potential benefit of therapy with BI 836858 is expected to outweigh the treatment-related risks.

## 3. DESCRIPTION OF DESIGN AND TRIAL POPULATION

#### 3.1 OVERALL TRIAL DESIGN AND PLAN

This trial will be performed in two separate patient populations: 1) Patients diagnosed with relapsed or refractory AML who have failed at least one prior line of therapy and 2) patients with AML who are in complete remission (CR) with a high risk to relapse. It will be performed in an open, non-randomized, 3+3 design followed by an expansion cohort. A cycle will comprise of 14 days.

For patients with refractory or relapsed AML, one cycle is 14 days with two administrations of BI 836858 (i.e. administrations on Days 1 and 8). Patients with clinical benefit, defined by the International Working Group (IWG) as having objective response (partial remission (PR) or complete remission (CR) or complete remission with incomplete blood recovery (CRi)) or subjective response (in the absence of objective response) after 8 administrations and who are tolerating the infusions, may continue until progressive disease (PD) and as long as neither patient nor Investigator requests treatment discontinuation.

<u>For AML patients in CR</u>, one cycle is 14 days with one administration of BI 836858 (i.e. administrations on Days 1) in Cycles 1, 2 and 3. From the 4<sup>th</sup> cycle onwards, patients will receive monthly (every second cycle) infusions of BI 836858 (i.e. 4<sup>th</sup> infusion on Cycle 5 Day 1, 5<sup>th</sup> infusion on Cycle 7 Day 1) for overall up to one year of treatment unless these patients relapse or infusions are not tolerated.

To determine separate MTDs for each patient population, cohort dose escalation will be conducted following the 3+3 design for the refractory or relapsed AML patients and the patients with AML in CR with high risk to relapse, respectively. The dose level will be escalated with each new cohort until at least one out of three patients of a cohort experiences a dose limiting toxicity (DLT; for definition see Section 5.2.1.1) during the first two cycles (DLT evaluation period). If exactly one out of the three patients of the cohort experiences a DLT, three additional patients will be treated at the same dose level. If none of the three additional patients experiences a DLT, then the cohort dose escalation will be continued by treating the next three patients at the next higher dose level. If at least two out of up to six patients at a dose level experience a DLT, the MTD has been exceeded and the dose will be deescalated until a dose level is reached in which at most one DLT out of six patients is observed (R01-0028). The MTD is defined as the dose of BI 836858 that is one dose cohort below the dose at which two or more out of six patients experienced DLT. At the maximum tolerated dose, no more than one patient out of six patients may experience DLT, i.e., the MTD is defined as the highest dose studied for which the incidence of dose-limiting toxicity is no more than 17% (i.e. 1/6 patients) during the first two cycles.

Patients are considered to have completed the first two cycles if they have reached end of cycle 2 and have received all planned administrations of BI 836858 (i.e. 4 administrations for patients with relapsed or refractory AML and 2 administrations for patients in CR).


However, for those patients who receive more than two cycles of BI 836858, all DLT occurring after end of cycle 2 will be taken into consideration for further development of BI 836858.

Table 3.1: 1 Table of action taken in response to DLTs

| Patients oxperiencing a | Number of patients in cohort | Action taken by Sponsor |
|---|---|---|
| experiencing a DLT | Colloit | |
| 0 | 3 | Open the next cohort |
| 1 | 3 | Add 3 additional patients (see below) at same dose level |
| 1 | 6 | If there are no new DLTs in additional 3 patients, open next cohort |
| 2 | 6 | If there is at least one new DLT in additional 3 patients, MTD is exceeded, expansion cohort opened at next lower dose level. |

During the dose escalation phase, each patient will receive up to 2 repeated treatment cycles before DLT assessment.

For both patient populations the dose is planned to be escalated in cohorts at pre-defined dose levels based on a multiplication factor of 2. The dose levels are 10 mg, 20 mg, 40 mg, 80 mg, 160 mg, and 320 mg as outlined in Section 4.1.3. However, for AML patients in CR, the dose escalation will start with the 40 mg dose cohort and follow the same dose escalation levels. Intermediate dose levels and dose levels higher than 320 mg may be investigated if agreed upon between Investigator and Sponsor.

After definition of the MTD, it is planned to enroll an expansion cohort of 12 patients to better characterize the safety of BI 836858. In case no MTD is reached up to the highest planned dose (e.g., 320 mg), 12 additional patients will be treated with each respective schedule at the-highest test dose (i.e., 320 mg) of BI 836858.

The primary analysis will take place when all patients from the cohort dose escalation and dose expansion cohorts have had a minimum of 4 cycles or have discontinued from the trial prior to reaching end of cycle 4 due to meeting the criteria for withdrawal as outlined in Section 3.3.4.1.

#### 3.1.1 Administrative structure of the trial

Boehringer Ingelheim is the Sponsor of this trial. The Coordinating Investigator will be participating Investigators will be physicians experienced and specialized in the treatment of AML and in the conduct of Phase I trials.

In regular telephone conferences between the participating Investigators and the Sponsor, there will be discussions of safety assessments, recommendations for cohort dose escalation, to reach a consensus on DLT, and whether to continue or modify the trial.

All safety laboratory analyses will be performed locally at each clinic site in the schedule outlined in the <u>Flow Charts</u>. All of the biomarker analyses will be performed at with the exception of cytokine analyses which will be performed in locations noted in <u>Section 5.6.3</u>.

# 3.2 DISCUSSION OF TRIAL DESIGN, INCLUDING THE CHOICE OF CONTROL GROUP

The primary objective of this trial is to determine the MTD for both patient populations separately. The most important secondary objective is to assess the safety of BI 836858. This can be achieved by an open label, single arm design without a control group.

Adult patients with refractory/relapsed AML are considered eligible for this trial. Relapsed AML is defined as recurrent disease after prior remission of any duration. Refractory disease is defined as failure to achieve remission to most recently administered therapy. Patients with primary refractory disease, defined as failure to achieve remission to initial therapy, are eligible. Typically patients with primary refractory disease are defined as refractory after failure of two cycles of intensive induction. Patients with failure of a single cycle of induction are eligible for this trial if they refuse to receive a second induction cycle or if they are not candidates for a second intensive induction cycle. Patients receiving hypomethylating agents as initial induction should receive at least two cycles of induction before designation as refractory.

AML patients in CR who have been initially diagnosed with non-favorable genetics have a very high risk to relapse. Eligible patients for this trial should either have received induction and consolidation treatment and are not candidates for allogeneic hematopoietic stem cell transplantation (e.g. no donor available, not eligible/fit enough) or have received allogeneic hematopoietic stem cell transplantation. For those patients no standard therapy to maintain the CR is currently available.

These AML patient groups were selected for inclusion in this trial, because these patients constitute groups with unfavourable prognosis for whom currently no satisfactory standard treatment exists.

The trial design will follow a 3+3 design with cohort dose escalation and de-escalation for both patient groups. Once the MTD has been defined, an expansion cohort of 12 patients is planned to be enrolled to better characterize the safety profile and tolerability of the MTD. In case no MTD is reached up to the highest planned dose (e.g., 320 mg), 12 additional patients will be treated with the respective schedule of the highest tested dose (e.g., 320 mg) of BI 836858. This trial design is accepted for hematology Phase I studies.

For patients with refractory or relapsed AML, the first efficacy assessment via bone marrow aspirate will be performed after 2 cycles (4 administrations). Subsequent disease assessment will be performed after 4 cycles (8 administrations) and at the discretion of the Investigator.

For AML patients in CR, disease status will be followed up on a regular basis with peripheral blood count and a bone marrow assessment will be performed if suspicion of relapse. Patients with a MRD marker will be followed up on this marker as well, however this is explorative.

Intra-patient dose escalation will be allowed for selected patients in case the next higher dose cohort is free of DLT and considered safe. This is not considered a safety risk because it will be restricted to patients who have tolerated at least three cycles of BI 836858 at the time of dose escalation and may offer a potential benefit to patients enrolled at a lower dose.

Each patient will be closely monitored for infusion-related reactions, as this is a potential side-effect for mAbs.

Safety assessments will be performed at all visits during the treatment phase.

The trial shall allow the investigation of BI 836858 in AML with regard to safety and the definition of the optimal dose for the future clinical development program in this disease.

#### 3.3 SELECTION OF TRIAL POPULATION

Approximately 50 patients with relapsed or refractory AML and about 35 AML patients in CR with high risk to relapse will be screened. Of these patients, approximately 36 with refractory or relapsed AML and approximately 27 patients with AML in CR with high risk to relapse will be included in this trial from a target of 5 sites. Each site will screen a target of about 10 patients.

A log of all patients included into the study (i.e. having given informed consent) will be maintained in the investigator site file (ISF) at the investigational site irrespective of whether they have been treated with investigational drug or not.

## 3.3.1 Main diagnosis for study entry

Patients with relapsed or refractory AML as defined according to the World Health Organization (WHO) criteria will be eligible for this trial (see Section 3.2),

#### **AND**

Patients with AML in CR with high risk to relapse will be eligible for this trial (see also Section 3.2). AML in CR with high risk to relapse is defined as follows:

a) AML patients with non-favorable genetics (according to European LeukemiaNet (ELN) classification) that are in CR after having received induction and consolidation chemotherapy and are not candidates for allogeneic hematopoietic stem cell transplantation (SCT) (e.g., no donor available, not eligible/fit enough)

or

b) AML patients with non-favorable genetics (according to ELN classification) that are in CR after allogeneic hematopoietic stem cell transplantation.

CR is defined as following: Morphologically leukemia free state (i.e. bone marrow with <5% blasts by morphologic criteria and no blasts with Auer rods, no evidence of extramedullary leukemia) and absolute neutrophil count  $\geq 1000 \ / \mu L$  and platelets  $\geq 100,000 \ / \mu L$ . However, for being eligible for this trial, patients in CR must **not** be independent of red blood cell transfusions.

#### 3.3.2 Inclusion criteria

- 1. Two patient populations: Patients with diagnosis of relapsed or refractory AML with at least one prior treatment for AML and patients with diagnosis of AML in CR with high risk to relapse.
- 2. <u>For patients with refractory or relapsed AML</u>: Expression of CD33 on more than 30% of bone marrow blasts per central laboratory assessment at the Ohio State University.

For AML patients in CR with high risk to relapse: Patients should have had a CD33 positive expression of bone marrow blasts at the time of initial AML diagnosis. No CD33 expression confirmation at screening is required.

- 3. Eastern Cooperative Oncology Group (ECOG) Performance Status ≤2. See Section 10.2
- 4. Age  $\geq$ 18 years.
- 5. Written informed consent which is consistent with International Conference on Harmonization Good Clinical Practice (ICH-GCP) guidelines and local legislation.

#### 3.3.3 Exclusion criteria

- 1. Patients with acute promyelocytic leukemia according to WHO definition
- 2. Patients with refractory or relapsed AML, >5,000 blasts in the peripheral blood.
- 3. Anti-leukemia therapy within two weeks before first treatment with BI 836858; however, parallel treatment with Hydroxyurea is allowed for patients with relapsed/refractory AML. (See Section 4.2.2.1)
- 4. Allogeneic stem cell transplantation within the last 28 days before first treatment with graft versus host disease requiring more than 20 mg of steroids per day. Steroid dosage must be stable within two weeks prior to start of treatment.
- 5. Patients who are candidates for allogeneic stem cell transplantation (for patients with refractory or relapsed AML).
- 6. Second malignancy currently requiring active therapy. However, patients with organ-confined prostate cancer with no evidence of recurrent or progressive

- disease based on prostate-specific antigen values are also eligible for this study if hormonal therapy has been initiated, or a radical prostatectomy or definitive radiotherapy has been performed.
- 7. Symptomatic central nervous system involvement (see Section 4.2.2)
- 8. Aspartate amino transferase (AST) or alanine amino transferase (ALT) greater than 2.5 times the upper limit of normal (ULN), or AST or ALT greater than 5 times the ULN for those with Gilbert syndrome.
- 9. Prothrombin time (PT) >1.5 x ULN for subjects not on therapeutic vitamin K antagonists (phenprocoumon, warfarin)
- 10. Bilirubin greater than 1.5 mg/dl (>26 μmol/L) unless elevation is thought to be due to hepatic infiltration by AML, Gilbert syndrome, or hemolysis.
- 11. Serum creatinine greater than 2.0 mg/dl
- 12. Known human immunodeficiency virus (HIV) infection or active hepatitis B virus or hepatitis C virus infection. Patients with any serological evidence of current or past hepatitis B exposure are to be excluded unless the serological findings are clearly due to vaccination
- 13. Concomitant intercurrent illness, or any condition which in the opinion of the Investigator, would compromise safe participation in the study, e.g. active severe infection, unstable angina pectoris, new onset of exacerbation of a cardiac arrhythmia
- 14. Psychiatric illness or social situation that would limit compliance with trial requirements
- 15. Concomitant therapy, which is considered relevant for the evaluation of the efficacy or safety of the trial drug (see Section 4.2.2)
- 16. Female patients of childbearing potential who are sexually active and unwilling to use a medically acceptable method of contraception during the trial and for 6 months after the last administration of BI 836858, i.e. combination of two forms of effective contraception (defined as hormonal contraception, intrauterine device, condom with spermicide, etc.). Subjects will be considered to be of childbearing potential unless surgically sterilized by hysterectomy, or bilateral tubal ligation/salpingectomy or post-menopausal for at least two years
- 17. Male patients with partners of childbearing potential who are unwilling to use condoms in combination with a second effective method of contraception (defined as hormonal contraception, intrauterine device, condom with spermicide, etc.) during the trial and for 6 months after the last administration of BI 836858
- 18. Pregnant or nursing female patients
- 19. Treatment with another investigational agent under the following conditions:
  - a) Within two weeks (for biologics 4 weeks or 5 half-lives, whichever is longer) of first administration of BI 836858; or
  - b) Patient has persistent toxicities from prior anti-leukemic therapies which are determined to be relevant by the Investigator.
  - c) Concomitant treatment with another investigational agent while participating in this trial.
- 20. Prior treatment with a CD33 antibody
- 21. Patient unable or unwilling to comply with the protocol.


28 Apr 2016

#### 3.3.4 Removal of patients from therapy or assessments

#### 3.3.4.1 Removal of individual patients

An individual patient is to be withdrawn from the trial if:

- The patient withdraws consent. Patients are free to discontinue their participation in this trial at any time without the need to justify the decision.
- The patient needs to take concomitant drugs which may interfere with the investigational product (please refer to Section 4.2.2).
- The patient is no longer able to participate for other medical reasons (e.g. adverse events unrelated to therapy or disease progression, concomitant diagnoses, pregnancy, surgery or administrative reasons). The Investigator may also stop a patient's participation if the patient is no longer able to attend trial visits.

A patient can be withdrawn from the trial after discussion between the Investigator and the Sponsor if eligibility criteria are violated and/or the patient fails to comply with the protocol.

All withdrawals will be documented and the reason for withdrawal recorded and discussed, as necessary, in the final report of the trial. As soon as a refractory or relapsed AML patient is withdrawn from the trial treatment, the end of active treatment (EOT) visit has to be performed if feasible. For patients with AML in CR, as soon as a patient is withdrawn from the trial treatment, the end of active treatment (EOT) visit and the End of Residual Effect Period (REP) visit (EoR visit) must be performed if feasible. Every effort should be made to follow-up with patients in case an adverse event (AE) is still ongoing at the time of withdrawal. If a patient is withdrawn from the trial due to consent withdrawal, no further visits will be completed and no further trial data will be collected. However, if information about survival status is available in the public domain, then the Investigator is requested to report this information in the eCRF.

A patient has to discontinue trial drug administration in case:

- A DLT occurs which does not recover to a degree that allows treatment continuation (see Section 4.1.4).
- Progressive disease (PD) or any other concomitant diagnosis/symptom develops resulting in an indication to start any other therapy for AML, including deterioration of general condition.

Patients not completing the first two cycles (with all planned BI 836858 administrations) for reasons other than DLT will be replaced.

## 3.3.4.2 Discontinuation of the trial by the sponsor

Boehringer Ingelheim reserves the right to discontinue the trial overall or at a particular trial site at any time for the following reasons:
Boehringer Ingelheim 28 Apr 2016 BI Trial No.: 1315.1

- 1. Violation of GCP, the Clinical Trial Protocol (CTP), or the contract by a trial site or Investigator, disturbing the appropriate conduct of the trial,
- 2. Emergence of any efficacy/safety information that could significantly affect continuation of the trial,
- 3. Failure to meet expected enrolment goals overall or at a particular trial site.
- 4. Any other administrative reasons, including discontinuation of the clinical development program with BI 836858.

The Investigator / the trial site will be reimbursed for reasonable expenses incurred in case of trial termination (except in case of the first reason).

## 4. TREATMENTS

#### 4.1 TREATMENTS TO BE ADMINISTERED

BI 836858 will be administered as rate-controlled intravenous infusion. In case a patient experiences an adverse event during the infusion, the duration of the infusion may be expanded until the use-by date and use-by time indicated on the label is reached. The actual duration of the infusion needs to be documented in the electronic case report form (eCRF) including actual start and end time, actual time points for interruption and restart of the infusion and the actual infusion rates.

Adverse events during the infusion will be thoroughly documented and characterized to allow differentiation between infusion-related reactions (<u>R10-4428</u>, <u>R10-4517</u>).

## 4.1.1 Identity of BI investigational product and comparator product

The characteristics of the test product are below.

• Substance (INN): BI 836858

• Pharmaceutical form: Solution for infusion after dilution

• Source: Boehringer Ingelheim Pharma GmbH & Co. KG

• Unit strength: 10 mg/mL (vials with 10mL)

• Daily dose: See <u>Section 4.1.3</u>

• Duration of use: Single administration every 7, 15, or 29 days

(depending on patient population)

• Route of administration: Intravenous

Posology: Rate controlled infusion

(Volume: 250 mL)

The first and second infusion will be started at a rate of 10 mL/h. The infusion rate should be increased every 30 (+/-10) minutes by 10 mL/h to a maximum of 80 mL/h as long as tolerated by the patient. Infusion should not exceed 8 hours. If considered safe by the Investigator, the stepwise increase of infusion rate during the third and subsequent infusions may be faster or steps may be omitted, but the maximum infusion rate must not exceed 120 mL/h. If symptoms of an infusion-related reaction occur, the infusion should be temporarily stopped. Upon recovery, it should be infused at 50% of the rate at which the reaction occurred and should not be dose escalated from this dose for at least 30 minutes. Lower rates may be selected if clinically indicated. Depending on the time of occurrence and the severity of the reaction, the investigator may consider administering additional supportive medication, e.g. corticosteroids. A stepwise re-increase of the infusion rate to a maximum of 80 mL/h is possible. For medical reasons, in case a patient experiences an adverse event during the infusion, the duration of the infusion may be expanded until the use-by date and use-by time indicated on the label is reached. The actual duration of the infusions and infusion steps need to be documented in the eCRF including actual start and end time, actual time points for interruption and restart of the infusion and the actual infusion rates.

hringer Ingelheim 28 Apr 2016


**Trial Protocol** 

## 4.1.2 Method of assigning patients to treatment groups

Not applicable. This is a single-arm, open-label, cohort dose escalation trial.

#### 4.1.3 Selection of doses in the trial

BI 836858 will be administered as a rate-controlled intravenous infusion every 7 days to refractory or relapsed AML patients.

For AML patients in CR, the first three administrations will be given every second week, on day 1 of Cycles 1, 2 and 3. From the 4<sup>th</sup> administration onwards, patients will receive monthly (every second cycle) infusions of BI 836858 (i.e. 4<sup>th</sup> infusion on Cycle 5 Day 1, 5<sup>th</sup> infusion on Cycle 7 Day 1...) for overall up to 12 months of treatment unless these patients relapse or infusions are not tolerated.

Patients with refractory or relapsed AML have a high medical need and a bad prognosis. To treat this patient population with a sub saturating dose is not warranted and therefore a starting dose close to the full saturation of all CD33 sites is chosen. The starting fixed dose of 10 mg which is a dose level expected to provide near to the full saturation of all CD33 sites at maximum measured plasma concentration (C<sub>max</sub>) based on estimated receptor occupancy (i.e. 94.3% estimated CD33 occupancy). For lintuzumab, a CD33 monoclonal antibody, in a Phase I trial no MTD was reached up to 8mg/kg/week (R11-1481). A fixed dose regimen was chosen instead of a dose per m² based a recent publication by Wang et al. The individual and population performance of body size-based and fixed dosing in adults were compared for 12 oncology approved mAbs (R10-6267). Although both dose regimens demonstrated similar performance, the fixed dose was recommended since it offered advantages in the ease of dose preparation and a lower chance of dosing errors.

For details please refer to the Investigator's Brochure, Section 5.3.6 (c02324887-03).

The dose is planned to be escalated in cohorts at pre-defined dose levels based on a multiplication factor of 2. The dose levels are 10 mg, 20 mg, 40 mg, 80 mg, 160 mg, and 320 mg. Intermediate dose levels and dose levels higher than 320 mg may be investigated if agreed upon between Investigator and Sponsor. In an ongoing Phase I study BI 836858 is administered to lower risk MDS patients every 14 days. In the 20 and 40 mg cohort no DLT occurred and the 80mg cohort is currently ongoing. The dose escalation in AML patients in CR will begin with infusions at the dose level of 40 mg. The dose will be escalated to the next pre-defined or intermediate dose levels as needed.

When a cohort dose escalation is to be performed, the data of all previous dose cohorts will be reviewed and discussed between the participating Investigators and the Sponsor. This assessment will determine if each patient population is able to continue treatment with BI 836858.

During the cohort dose escalation phase, enrolment into the first dose cohort (10 mg) will be allowed at the earliest 7 days after the first administration of BI 836858 between patient 1


and 2 and subsequently between patient 2 and 3. In case the 10 mg cohort has to be expanded to 6 patients, a one week observation period must be followed between the first administration of BI 836858 and the start of the subsequent patient. For subsequent cohorts (i.e., 20 mg, 40 mg, 80 mg, 160 mg, and 320 mg), consecutive screening is allowed; however, there has to be an interval of at least 3 days between the 1<sup>st</sup> administration of BI 836858 for each patient.

Enrolment into the next higher dose cohort is allowed after the previous dose cohort was found to be safe for the initial administration for all patients in this cohort (e.g. at least 28 days after the first administration of drug in the last patient entered into the cohort).

Once the MTD for one of the patient populations is defined, a dose for treatment of the expansion cohort in this patient population will be determined, which will not exceed the MTD. In case no MTD is reached up to the highest tested dose (e.g. 320 mg), 12 additional patients will be treated with the respective schedule of the highest tested dose (e.g. 320 mg) of BI 836858 in the expansion cohort. During treatment of the expansion cohort, new patients may be enrolled at any time.

Table 4.1.3: 1 Entry of patients into trial, by cohort

| Cohort | Day first patient in cohort receives infusion | Earliest day<br>next patient can<br>be enrolled |
|---|---|---|
| 10 mg* | Day 1 | Day 8 |
| All other dose levels in cohort** dose escalation | Day 1 | Day 4 |
| Dose Expansion | Day 1 | Any time |

<sup>\*</sup> a one week observation period must be followed between the first administration of BI 836858 and the start of the subsequent patient - for all patients with refractory or relapsed AML in the 10 mg cohort \*\*This entry schedule also applies to AML patients in CR, starting at 40 mg cohort.

#### 4.1.4 Drug assignment and administration of doses for each patient

Prior to inclusion of a new patient during the cohort dose escalation phase, the Investigator has to confirm the actual dose tier of BI 836858 for the patient with the Sponsor who oversees the cohort dose escalation steps and the safety data of patients from all trial sites. BI 836858 will be administered as an intravenous infusion under the supervision of the Investigator or designated personnel.

BI 836858 may be administered at any time during the day. However, to it is recommended to start the infusion during the morning hours.

Trial Protocol 

<u>For refractory or relapsed AML patients</u>: BI 836858 will be administered as weekly i.v. infusions in 14-day cycles (i.e., Days 1 and 8; 2 infusions per cycle).

<u>For AML patients in CR</u>: the first three administrations will be given once every second week on day one of 14-day Cycles 1, 2 and 3 (i.e., Days 1, 15 and 29). From the 4<sup>th</sup> administration onwards, patients will receive monthly (every second cycle) infusions of BI 836858 (i.e. 4<sup>th</sup> administration on Cycle 5 Day 1, 5<sup>th</sup> administration on Cycle 7 Day 1 ...) for overall up to 12 months of treatment.

#### Premedication

Premedication to prevent infusion-related reactions is obligatory 30 minutes (up to 120 min before start of administration of BI 836858 is permissible) prior to the first three administrations of BI 836858, unless a contraindication for premedication exists, and should include:

- Acetaminophen/Paracetamol 650 mg 1000 mg p.o., or equivalent
- Antihistamine p.o. or i.v., equivalent to Diphenhydramine 50 mg i.v.
- Glucocorticoid i.v., equivalent to prednisolone 100 mg

## For patients with refractory or relapsed AML:

If BI 836858 has been well tolerated without signs of infusion-related reactions in the first administration, glucocorticoid premedication may be reduced to a dose equivalent to 50 mg prednisolone for the second through fourth administrations, and in case this is well tolerated reduce the steroids with the 5th infusion (25 mg with the 5<sup>th</sup> and 0 mg with the 6<sup>th</sup> infusion.)

#### For AML patients in CR:

If BI 836858 has been well tolerated without signs of infusion-related reactions in the first administration, glucocorticoid premedication may be reduced to a dose equivalent to 50 mg prednisolone for the second administration, and in case this is well tolerated steroids can be omitted with the 3rd infusion.

For <u>both</u> patient populations, however, in case an administration of BI 836858 was not well tolerated, the premedication with prednisolone can be re-escalated up to 100 mg.

#### Retreatment

Before the next administration of BI 836858, adverse events and safety laboratory will be assessed. To continue treatment with further administrations, all of the following criteria must be met:

#### Refractory or relapsed AML patients

Neutrophils  $\geq$ 500 /µL (0.5 x 10<sup>9</sup>/L) and platelets  $\geq$ 25,000 /µL (25 x 10<sup>9</sup>/L), unless CTCAE Grade 4 neutropenia or thrombocytopenia was preexistent prior to trial entry. Patients with active leukemia who go from Grade 3 neutropenia to Grade 4 neutropenia after treatment may continue on study provided there is no evidence of infection or febrile neutropenia. Patients with active leukemia who go from

Grade 3 to Grade 4 thrombocytopenia after treatment may continue on study provided that post-transfusion platelet count is at least  $20,000/\mu L$  before therapy is given.

(2) Acceptable tolerability (in case of an AE at the planned start of a further administration, patients may continue therapy only after recovery to a level which would allow further therapy, i.e. CTCAE grade 1 or pre-treatment value); no febrile neutropenia (≥38.5°C and ANC <1000/µL) and no uncontrolled infection. Patients who do not meet these criteria for further therapy should be discussed with the TCM and/or the Coordinating Investigator and may be eligible to continue if the toxicity is not clinically significant.

## AML patients in CR

- (1) Neutrophils  $\geq 750 / \mu L (0.75 \times 10^9 / L)$  and platelets  $\geq 50,000 / \mu L (50 \times 10^9 / L)$ .
- (2) Acceptable tolerability (in case of an AE at the planned start of a further administration, patients may continue therapy only after recovery to a level which would allow further therapy, i.e. CTCAE grade 1 or baseline value.)
- (3) Patients with GvHD, with a CTCAE grade 1 or 2 and taking steroids, may continue further administration. GvHD patients with a steroid-refractory (≥2 mg/Kg) CTCAE grade 3 or higher, independent of receiving steroids, should be discontinued from study.

In case criteria 1 and 2 are not fulfilled, blood counts and/or the adverse event should be re-evaluated for up to three weeks. In case of a treatment delay, the Sponsor must be notified. If criterion 1 is not fulfilled and the patient has <5% blasts in the bone marrow, absence of myelodysplastic changes, and/or absence of evidence of disease by flow cytometry in the bone marrow then no further treatment should be administered until discussion with the Sponsor.

Administration of the trial drug has to be stopped temporarily in case of a DLT (see Section 5.2.1.1). Patients may continue therapy only after recovery from the DLT to a CTCAE level which allows further therapy based on Investigator assessment and only with a reduced dose of BI 836858. The new dose of BI 836858 must be finally agreed on between the Sponsor and the Investigator. The reduced dose will be valid for all following treatment cycles in the individual patient. A reduction of the dose will be allowed only once for an individual patient during the whole trial. In case a patient experiences a second episode of DLT with the reduced BI 836858 dose, the treatment has to be permanently discontinued. Likewise, treatment has to be discontinued in case the DLT is not reversible.

## *Intra-patient dose escalation*

Intra-patient dose escalation may be considered in agreement between investigator and sponsor for selected patients. It is restricted to patients who have received at least 3 treatment cycles and tolerate the treatment well at the time of dose escalation. Intra-patient dose escalation can only be performed at a time when the next higher dose cohort has been

reviewed and considered safe by the sponsor and investigators. The dose escalation step is limited to the dose which has been administered to the next higher cohort. In addition, after the first dose at the higher dose level, patients have to be monitored for at least 24 hours after the end of the infusion, including safety laboratory 24 hours after the first administration of the escalated dose of BI 836858.

A log of all patients enrolled into the study (i.e. having given informed consent) will be maintained in the Investigator Site File (ISF) at the investigational site irrespective of whether they have been treated with investigational drug or not.

## 4.1.5 Blinding and procedures for unblinding

## 4.1.5.1 Blinding

This Phase I trial will be performed according to an open label, single arm design. It will recruit two separate patient populations: 1) Patients with relapsed and refractory AML and active disease; and 2) AML patients in CR with high risk to relapse. This trial will be handled in an open fashion by the Sponsor throughout, i.e. also for the purpose of data cleaning and preparation of the analysis. The eCRF will contain information on the treatment and the dose.

## 4.1.5.2 Procedures for emergency unblinding

Not applicable.

## 4.1.6 Packaging, labelling, and re-supply

BI 836858 will be supplied in 10 mL vials containing 100 mg BI 836858. For details of packaging and the description of the label, refer to the ISF. Medication will be delivered to the Investigator's pharmacy where the total dose per patient will be prepared upon request from the Investigator.

For preparation of BI 836858 infusion solution, the content of the vial of BI 836858 will be diluted in 0.9% sodium chloride. The content of several vials may be needed for administration of the requested dose. For further details, please refer to the instructions included in the ISF. The full volume of the diluted compound will be 250 mL.

## 4.1.7 Storage conditions

BI 836858 has to be stored in a limited access area at the temperature indicated on the trial drug label - stored in a refrigerator 36-46°F (2-8°C); do not freeze. If the storage conditions are found to be outside the specified range, immediately contact the local clinical monitor (CML) as provided in the list of contacts. For more details on BI 836858, please refer to the Investigator's Brochure (IB) and the ISF.

## 4.1.8 Drug accountability

Drug supplies of BI 836858, which will be provided by the Sponsor or a Clinical Research Organization (CRO) appointed by the Sponsor, must be kept in a secure, limited access storage area under the storage conditions defined by the Sponsor. A temperature log must be maintained to make certain that the drug supplies are stored at the correct temperature.

Each Investigator and/or pharmacist will receive the investigational drugs delivered by the Sponsor when the following requirements are fulfilled:

- approval of the study protocol by the IRB / ethics committee,
- availability of a signed and dated clinical trial contract between the sponsor and the Head of Trial Centre.
- approval/notification of the regulatory authority, e.g. competent authority,
- availability of the curriculum vitae of the principal Investigator,
- availability of a signed and dated CTP or immediately imminent signing of the CTP,
- availability of the proof of a medical licence for the principal investigator,
- availability of the Form 1572.

These records will include dates, quantities, batch/serial numbers, expiry ('use by') dates, and the unique code numbers assigned to the investigational product(s) and trial patients. The Investigator and/or pharmacist must maintain records of the product's delivery to the trial site, the inventory at the site, the use for each patient, and the return to the Sponsor or alternative disposition of unused product. The Investigator/pharmacist will maintain records that document adequately that the patients were provided these doses specified by the CTP and reconcile all investigational product received from the Sponsor. At the time of return to the sponsor, the investigator must verify that all unused or partially used drug supplies have been returned by the clinical trial patient and that no remaining supplies are in the investigator's possession.

## 4.2 CONCOMITANT THERAPY, RESTRICTIONS, AND RESCUE TREATMENT

## 4.2.1 Rescue medication, emergency procedures, and additional treatments

Rescue medication to reverse the action of BI 836858 is not available. Potential side effects of BI 836858 have to be treated symptomatically. Patients should receive supportive care according to the local guidelines regarding treatment of infusion-related reactions, blood product support, antibiotics, antivirals, analgesics, skin and mouth care, etc. The use of growth factors such as granulocyte colony stimulating factor (G-CSF) will be allowed, but growth factors should be avoided during the first 2 cycles for better assessment of safety and response parameters.

Anti- bacterial and fungal prophylaxis should be given according to local standards or available guidelines.

Boehringer Ingelheim BI Trial No.: 1315.1 Doc. No.: c02543230-04 28 Apr 2016


All concomitant non-anti-leukemia therapies to provide adequate care may be given as clinically necessary. All concomitant treatments will be recorded in the eCRF except for vitamins and nutrient supplements. Trade name, indication and dates of administration of concomitant therapies will be documented. For parenteral nutrition during the trial, the components need not be specified in detail. It should be indicated as 'parenteral nutrition'. If a patient needs anesthesia, it will be sufficient to indicate 'anesthesia' without specifying the details.

**Trial Protocol** 

Concomitant therapy will be recorded in the eCRF during the screening and treatment period, starting at the date of signature of informed consent, and ending at the EOT-visit. After the EOT-visit, only concomitant therapy indicated for treatment of an adverse event needs to be reported.

## 4.2.2 Restrictions

## 4.2.2.1 Restrictions regarding concomitant treatment

Prior anti-leukemia therapy must have been discontinued at least two weeks before the first administration of the trial drug (Hydroxyurea may be given during study participation) and the patient must have recovered from all clinically relevant reversible toxicities as determined by the investigator. A time interval of at least 2 weeks (four weeks for biologics) must have elapsed from the last administration of any other investigational treatment for AML to the first administration of BI 836858.

For peripheral blood blast control, as this may correlate with the risk of occurrence of infusion related symptoms, hydroxyurea will be allowed (maximum dose of hydroxyurea 3gm daily) before and during study participation. Blasts must be  $\leq 5,000/\mu l$  at start of each administration of BI 836858.

No other anti-neoplastic therapy concomitantly is allowed.

Short term glucocorticoid medications may be used up to 20 mg per/day continuously are allowed (see exclusion criterion 4) and up to 2 mg/kg bodyweight for short term. All other indications for steroids have to be discussed and agreed upon between Investigator and Sponsor.

Intrathecal treatment to control symptoms associated with central nervous system (CNS) involvement is allowed but must be discussed and agreed upon between Investigator and Sponsor. All concomitant therapy will be recorded in the eCRF.

## 4.2.2.2 Restrictions on diet and life style

No restrictions apply with regard to diet or life style.

Boehringer Ingelheim
28 Apr 2016
BI Trial No.: 1315.1

## 4.3 TREATMENT COMPLIANCE

BI 836858 will be administered as a single intravenous infusion under supervision of the Investigator or dedicated clinic personnel. Compliance may also be verified by pharmacokinetic assessment. Any discrepancies will be explained in the eCRF by the Investigator or designee.

## 5. VARIABLES AND THEIR ASSESSMENT

### 5.1 EFFICACY – PHARMACODYNAMICS

## **5.1.1 Endpoints of efficacy**

The efficacy endpoints will be assessed at the time points specified in the <u>Flow Charts</u>. Efficacy endpoints will be secondary in this trial.

Secondary endpoints of efficacy are:

## For patients with refractory or relapsed AML:

- Best overall response according to International Working Group (IWG) criteria (please see Section 5.1.2.3) (R06-0452)
- Progression free survival
- Time to treatment failure

## For AML patients in CR with high risk to relapse:

- Progression free survival
- Time to treatment failure

## 5.1.2 Assessment of efficacy

### 5.1.2.3 Assessment and definition of best overall response

For patients with refractory or relapsed AML, response will be assessed according to the criteria from the IWG based on laboratory data from the peripheral blood, bone marrow examination, clinical examination (at the end of each cycle), at the evaluation for further treatment-visit and the EOT-visit. Bone marrow examination will be performed before the Cycle 3 and Cycle 5 (5th and 9th administration of BI 836858) (i.e., BM performed on Day 1 (+/-1) of cycles 3 and 5 and treatment started on Day 1 (up to +3) of cycles 3 and 5) and at the discretion of the Investigator, e.g. in case clinical and laboratory examinations of peripheral blood demonstrate that a CR has been achieved, or for assessment of persistent neutropenia, anemia or thrombocytopenia.

For AML patients in CR, response will be assessed clinically and in the peripheral blood (on Day 1 of each cycle). In the case of suspected relapse based on peripheral blood counts a bone marrow examination will be performed.

## Assessment and definition of best overall response

Response will be evaluated according to the following criteria (modified from the IWG criteria, R06-0452):

## • Complete remission (CR)

Morphologically leukemia free state (i.e. bone marrow with <5% blasts by morphologic criteria and no blasts with Auer rods, no evidence of extramedullary leukemia) and absolute neutrophil count  $\geq 1000~\mu$ L and platelets  $\geq 100,000~\mu$ L. Patient must be independent of transfusions (no transfusion for 1 week prior to the assessment).

• Complete remission with incomplete blood count recovery (CRi)

All of the above criteria for CR must be met, except that absolute neutrophils  $<\!1000~/\mu L$  or platelets  $<\!100,\!000~/\mu L$  in the blood.

• Partial remission (PR)

All of the criteria for CR must be met, except that leukemic blasts in the bone marrow may range from 5 to 25% as long as the count has decreased by at least 50% from pre-study treatment, or <5% blasts in the presence of Auer rods or abnormal morphology.

• Stable disease (SD)

Patient alive with no CR, CRi, PR or PD.

## • Treatment failure (TF)

Patient survives ≥7 days following completion of initial 2 treatment cycles (e.g. 28 days) with persistent leukemia in the last peripheral blood smear or bone marrow (>25% blasts), or with persistent extramedullary disease, but without further clinical deterioration due to leukemia or increase of blast population in the bone marrow or peripheral blood.

Resistant disease: Patient survives  $\geq 7$  days post-course of treatment; persistent leukemia in blood or bone marrow.

Aplasia: Patient survives ≥7 days post-course of treatment; death while cytopenic, with aplastic bone marrow

Indeterminate cause: Patients who die < 7 days post therapy. Patients who die > 7 days post therapy with no peripheral blood blasts, but no bone marrow examination. Patients who do not complete the first course of therapy.

Morphologic relapse (recurrence): Reappearance of blasts post-CR or CRi in peripheral blood or bone marrow. That is, bone marrow leukemic blasts  $\geq 5\%$  or reappearance of blasts in the blood not attributable to any other cause (e.g. bone marrow regeneration), or development of extramedullary disease.

## • Progressive disease (PD)

Patient survives ≥7 days following completion of initial 2 treatment cycles (e.g. 28 days) with increase of blast population in the bone marrow or peripheral blood by >50% or aggravation or new development of extramedullary disease or further deterioration or death due to leukemia. Patients with a global deterioration of health status requiring discontinuation of treatment without objective evidence of PD at that time should be classified as having 'clinically progressive disease'. Every effort should be made to document the objective PD even after discontinuation of treatment.

## Definition of best overall response

Best overall response is defined as the best overall response (CR, CRi, PR, TF, PD or not evaluable in this order) recorded since first administration of BI 836858.

## 5.1.2.4 Progression free survival (PFS)

- PFS is defined as the time from first treatment with BI 836858 until disease progression, relapse or death.
- The date of progression/relapse will be the earliest of the dates of the disease assessment (blood sample, bone marrow sample, or clinical assessment) in which the

**Boehringer Ingelheim BI Trial No.: 1315.1** Doc. No.: c02543230-04 **Trial Protocol** 

28 Apr 2016

progression/relapse was observed. For patients who did not progress, relapse, or die, PFS will be censored at the date of last disease assessment.


#### Time to treatment failure (TTF) 5.1.2.5

Some patients will receive the next line of therapy, although no formal PD may be diagnosed at the time when the next treatment is indicated according to Investigator assessment. In addition to PFS, the TTF will be calculated.

- TTF is defined as the time from first treatment with BI 836858 until objective disease progression, relapse or death or start of next AML therapy.
- The date of progression/relapse will be the earliest of the dates of the disease assessment (blood sample, bone marrow sample, or clinical assessment) in which the progression/relapse was observed. For patients who did not progress, relapse, die, or receive next AML therapy TTF will be censored at the date of last disease assessment.


#### 5.2 SAFETY

## 5.2.1 Endpoints of safety

Primary endpoints:

- Maximum tolerated dose (MTD)
- Number of patients with Dose Limiting Toxicity (DLT) during the MTD evaluation period:
  - For patients with refractory or relapsed AML, the first two cycles (i.e. patient has received at least 4 administrations of BI 836858 and reached end of cycle 2).
  - For AML patients in CR with high risk to relapse, the first two cycles (i.e. patient has received at least 2 administrations of BI 836858 and reached end of cycle 2).

As this trial is the first in human use of BI 836858, the primary objective is to determine the MTD of BI 836858 and assess the safety of the drug in humans. For details on determination of MTD, please refer to Section 3.1, Section 5.2.1.1 and Section 7.3.1.

The safety of BI 836858 will be assessed by a descriptive analysis of incidence and intensity of adverse events (AE) graded according to the CTCAE version 4.0, the incidence of DLT, laboratory data and results of physical examination.

The Sponsor will review the safety data with the participating Investigators at regular intervals and as ad hoc if needed.

The safety endpoints will be assessed in a descriptive way without confirmatory analyses.

## 5.2.1.1 Dose limiting toxicity (DLT) for refractory or relapsed AML patients

DLT is defined as any non-disease-related non-hematological AE of CTCAE grade 3 or higher. Expected non-hematological disease related AE's such as complications resulting from haematological AEs include:

- bleeding and complications from bleeding due to thrombocytopenia as defined by the investigator
- infection and complications from infections due to neutropenia as defined by the investigator

• constitutional symptoms due to anemia as defined by the investigator

Infusion-related reactions (IRRs, CTCAE grade 3 or higher) associated with the administration of BI 836858 should be reported as Adverse Event of Special Interest (AESI, refer to Section 5.2.2.1), but will not be regarded as a DLT. The exception is anaphylaxis which occurs despite premedication with glucocorticoid or which does not resolve with glucocorticoid (i.e. such cases of anaphylaxis will be regarded as a DLT).

Infection will not constitute a DLT unless it is felt that the infection resulted from unexpectedly complicated myelosuppression; degree of severity and/or duration as assessed by the Investigator.

Hematological AEs, e.g. neutropenia, thrombocytopenia and anemia are frequently pre-existing in AML patients and are therefore AEs not considered as DLT. Failure to recover neutrophil count (ANC>500/uL) or platelet count (>25000/uL) at the first bone marrow evaluation after 2 cycles of BI 836858 in patients with < 5% blasts in the bone marrow, absence of myelodysplastic changes, and/or absence of evidence of disease by flow cytometry in the bone marrow will be considered a DLT. For patients with  $\geq$  5% blasts, myelodysplastic changes, or evidence of disease by flow cytometry/cytogenetics, failure to recover neutrophil or platelet count may not be considered DLT as this could be the result of persistent disease.

Patients who have not completed at least 4 administrations (2 cycles) of BI 836858 due to BI 836858 related toxicity will be considered as a DLT.

## 5.2.1.2 Dose limiting toxicity (DLT) for AML patients in CR

DLT is defined as any non-disease-related AE of CTCAE grade 3 or higher. Patients in remission are not expected to have disease-related AEs. In case of any hematological AE of CTCAE grade 3 or higher, relapse of AML has to be excluded. Infusion-related reactions (IRRs) associated with the administration of BI 836858 should be reported as Adverse Events of Special Interest (AESI, refer to Section 5.2.2.1), but will not be regarded as a DLT. The exception is anaphylaxis which occurs despite premedication with glucocorticoid or which does not resolve with glucocorticoid (i.e. such cases of anaphylaxis will be regarded as a DLT).

Occurrence of and/or worsening of GvHD will not be considered as a DLT; however, these cases will be reviewed carefully during the safety assessment meetings.

AML patients in CR who have not completed at least 2 administrations (2 cycles) of BI 836858 due to BI 836858 related toxicity will be considered as a DLT.

Once each patient of a cohort has completed 2 treatment cycles of BI 836858 all available safety data will be reviewed by the Sponsor, Coordinating Investigator and other participating Investigators who enrolled at least one patient. Safety data will be discussed via a


teleconference, initiated by Sponsor, to reach a consensus on DLT, in order to allow dose escalation, cohort expansion or suspension of further dose escalation.

All DLTs occurring at any time will be reported as an adverse event of special interest (AESI, see Sections 5.2.2.1 for definitions and 5.2.2.2 for reporting requirements).

### 5.2.2 Assessment of adverse events

### 5.2.2.1 Definitions of AEs

## Adverse event

An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation subject administered a medicinal product and which does not necessarily have to have a causal relationship with this treatment.

An AE can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.

## Adverse reaction

An adverse reaction is defined as a response to a medicinal product which is noxious and unintended. Response in this context means that a causal relationship between a medicinal product and an adverse event is at least a reasonable possibility. Adverse reactions may arise from use of the product within or outside the terms of the marketing authorisation or from occupational exposure. Conditions of use outside the marketing authorization include off-label use, overdose, misuse, abuse and medication errors.

## Serious adverse event

A serious adverse event (SAE) is defined as any AE which:

- results in death,
- is life-threatening, this refers to an event in which the patient was at risk of death at the time of the event; it does not refer to an event that hypothetically might have caused death if more severe.
- requires inpatient hospitalisation or
- prolongation of existing hospitalisation,
- results in persistent or significant disability or incapacity, or
- is a congenital anomaly / birth defect, or
- is to be deemed serious for any other reason if it is an important medical event when based upon appropriate medical judgment which may jeopardise the patient and may require medical or surgical intervention to prevent one of the other outcomes listed in the above definitions.

Medical and scientific judgement should be exercised in deciding whether other situations should be considered serious reactions, such as important medical events that might not be

Trial Protocol 

immediately life threatening or result in death or hospitalisation but might jeopardise the patient or might require intervention to prevent one of the other outcomes listed above. Examples of such events are intensive treatment in an emergency room or at home for allergic bronchospasm, blood dyscrasias or convulsions that do not result in hospitalisation or development of dependency or abuse. Any suspected transmission via a medicinal product of an infectious agent is also considered a serious adverse reaction.

## AEs considered "Always Serious"

Every new occurrence of cancer of new histology must be reported as a serious event regardless of the duration between discontinuation of the drug and the occurrence of the cancer.

Cancers of new histology and exacerbations of existing cancer must be reported as a serious event regardless of the duration between discontinuation of the drug and the occurrence of the cancer.

In accordance with the European Medicines Agency initiative on Important Medical Events, Boehringer Ingelheim has set up a list of further AEs, which by their nature, can always be considered to be "serious" even though they may not have met the criteria of an SAE as given above.

The latest list of "Always Serious AEs" can be found in the RDC system. A copy of the latest list of "Always Serious AEs" will be provided to you upon request. These events should always be reported as SAEs as described above.

## Adverse events of special interest (AESIs)

The term AESI relates to any specific AE that has been identified at the project level as being of particular concern for prospective safety monitoring and safety assessment within this trial, e.g. the potential for AEs based on knowledge from other compounds in the same class. AESI need to be reported to the sponsor's Pharmacovigilance Department within the same timeframe that applies to SAE, please see above.

The following are considered as AESIs:

- infusion-related reactions (CTCAE grade 3 or higher),
- any event that qualifies for DLT, and
- hepatic injury (DILI).

### Hepatic injury

A hepatic injury (DILI) is defined by the following alterations of hepatic laboratory parameters:

- an elevation of AST and/or ALT  $\geq$ 3 fold ULN combined with an elevation of total bilirubin  $\geq$ 2 fold ULN measured in the same blood draw sample, and/or
- marked peak aminotransferase (ALT, and/or AST) elevations ≥10 fold ULN


These lab findings constitute a hepatic injury alert and the patients showing these lab abnormalities need to be followed up according to the "DILI checklist" provided in the ISF. In case of clinical symptoms of hepatic injury (icterus, unexplained encephalopathy, unexplained coagulopathy, right upper quadrant abdominal pain, etc.) without lab results (ALT, AST, total bilirubin) available, the Investigator should make sure these parameters are analysed, if necessary in an unscheduled blood test. Should the results meet the criteria of hepatic injury alert, the procedures described in the DILI checklist should be followed

## Intensity of AEs

The intensity of adverse events should be classified and recorded in the CRF according to the Common Terminology Criteria for Adverse Events (CTCAE, version 4.0, <u>R09-2850</u>).

## Causal relationship of AEs

The definition of an adverse reaction implies at least a reasonable possibility of a causal relationship between a suspected medicinal product and an adverse event. An adverse reaction, in contrast to an adverse event, is characterised by the fact that a causal relationship between a medicinal product and an occurrence is suspected.

Medical judgment should be used to determine the relationship, considering all relevant factors, including pattern of reaction, temporal relationship, de-challenge or re-challenge, confounding factors such as concomitant medication, concomitant diseases and relevant history.

Arguments that may suggest that there is a reasonable possibility of a causal relationship could be:

- The event is consistent with the known pharmacology of the drug
- The event is known to be caused by or attributed to the drug class.
- A plausible time to onset of the event relative to the time of drug exposure.
- Evidence that the event is reproducible when the drug is re-introduced
- No medically sound alternative aetiologies that could explain the event (e.g. preexisting or concomitant diseases, or co-medications).
- The event is typically drug-related and infrequent in the general population not exposed to drugs (e.g. Stevens-Johnson syndrome).
- An indication of dose-response (i.e. greater effect size if the dose is increased, smaller effect size if dose is diminished).

Arguments that may suggest that there is no reasonable possibility of a causal relationship could be:

- No plausible time to onset of the event relative to the time of drug exposure is evident (e.g. pre-treatment cases, diagnosis of cancer or chronic disease within days / weeks of drug administration; an allergic reaction weeks after discontinuation of the drug concerned)
- Continuation of the event despite the withdrawal of the medication, taking into account the pharmacological properties of the compound (e.g. after 5 half-lives). Of note, this criterion may not be applicable to events whose time course is prolonged despite removing the original trigger.

0-04 Trial Protocol 

- Additional arguments amongst those stated before, like alternative explanation (e.g. situations where other drugs or underlying diseases appear to provide a more likely explanation for the observed event than the drug concerned).
- Disappearance of the event even though the study drug treatment continues or remains unchanged.

## 5.2.2.2 Adverse event collection and reporting

#### **AE Collection**

The Investigator shall maintain and keep detailed records of all AEs in their patient files. The following must be collected and documented on the appropriate CRF(s) by the Investigator:

• From signing the informed consent onwards through the Residual Effect Period (REP), until individual patient's end of trial:

All AEs (serious and non-serious) and all AESIs.

- However, if an individual patient discontinues trial medication prematurely but stays in the trial (i.e. if further visits incl. telephone visits, or vital status assessments are planned) from then on and until the individual patient's end of the trial the Investigator must report related SAEs and related AESIs.
- After the individual patient's end of trial:

The Investigator does not need to actively monitor the patient for AEs but should only report relevant SAEs and relevant AESIs of which the Investigator may become aware of.

The rules for Adverse Event Reporting exemptions (see below in paragraph "Exemptions to (S)AE Reporting") still apply.




The REP is defined as 30 days after the last trial medication application. All AEs which occurred through the treatment phase and throughout the REP will be considered as "on treatment," please see <u>Section 7.3.3</u>. Events which occurred after the REP will be considered as "post-treatment" events.

## AE reporting to sponsor and timelines

The Investigator must report SAEs, AESIs, and non-serious AEs which are relevant for the reported SAE or AESI, on the BI SAE form via fax immediately (within 24 hours) to the sponsor's unique entry point (country specific contact details will be provided in the ISF). The same timeline applies if follow-up information becomes available. In specific occasions the Investigator could inform the sponsor upfront via telephone. This does not replace the requirement to complete and fax the BI SAE form.

With receipt of any further information to these events, a follow-up SAE form has to be provided. For follow-up information the same rules and timeline apply as for initial information.

## Information required

For each AE, the Investigator should provide the information requested on the appropriate CRF pages and the BI SAE form. The Investigator should determine the causal relationship to the trial medication and any possible interactions between the investigational drug(s) and a Non-Investigational Medicinal Product (NIMP) / Auxiliary Medicinal Product (AMP).

The following should also be recorded as an (S)AE in the CRF and SAE form (if applicable):

- Worsening of the underlying disease or of other pre-existing conditions
- Changes in vital signs, ECG, physical examination and laboratory test results, if they are judged clinically relevant by the Investigator.

If such abnormalities already pre-exist prior trial inclusion they will be considered as baseline conditions.

All (S)AEs, including those persisting after individual patient's end of trial must be followed up until they have resolved, have been sufficiently characterised, or no further information can be obtained.

### Pregnancy

In rare cases pregnancy may occur in a clinical trial. Once a patient has been enrolled into this clinical trial and has taken trial medication, the Investigator must report immediately (within 24 h) a potential drug exposure during pregnancy (DEDP) in a female patient or in a partner to a male patient to the sponsor's unique entry point (country-specific contact details will be provided in the ISF). The Pregnancy Monitoring Form for Clinical Trials (Part A) should be used.

The outcome of the pregnancy associated with the drug exposure during pregnancy must be followed up and reported to the sponsor's unique entry point on the Pregnancy Monitoring Form for Clinical Trials (Part B).

As pregnancy itself is not to be reported as an AE, in the absence of an accompanying SAE, only the Pregnancy Monitoring Form for Clinical Trials and not the SAE form is to be completed. If there is an SAE associated with the pregnancy then the SAE has to be reported on the SAE form in addition.

The ISF will contain the Pregnancy Monitoring Form for Clinical Trials (Part A and B).

### Exemptions to (S)AE Reporting

Disease Progression in oncology trials is a study endpoint for analysis of efficacy, and as such is exempted from being reported as an SAE. Progression of the patient's underlying malignancy will be recorded on the appropriate pages of the eCRF as part of efficacy data collection only and will not be reported on the SAE Form. It will therefore not be entered in the safety database (Adverse Reactions Information System global, ARISg) and hence not get expeditiously reported. Death due to disease progression is also to be recorded on the appropriate eCRF page and not on the SAE Form.

Examples of exempted events of PD may be:

- Progression of underlying malignancy (Progressive disease [PD]): if PD is clearly consistent with the suspected progression of AML as defined by the respective response criteria.
- Hospitalization/Procedures due solely to the progression of underlying malignancy (PD)
- Clinical symptoms and/or signs of progression (without confirmation by objective criteria e.g. imaging, clinical measurement): If the symptom can exclusively be determined to be due to the progression of the underlying malignancy and does meet the expected pattern of progression for the disease under study.

However, when there is evidence suggesting a causal relationship between the trial drug and the progression of the underlying malignancy, the event must be reported as an (S)AE on the SAE Form and on the eCRF.

## **5.2.3** Assessment of safety laboratory parameters

## 5.2.3.1 General safety laboratory parameters

Blood samples and urine have to be collected at the time points specified in the <u>Flow Charts</u>. Safety laboratory examinations will include hematology, biochemistry, coagulation and qualitative urine analysis:

Hematology Hemoglobin, white blood cell count (WBC) with differential,

platelets (PLT)

Reticulocytes have to be measured only at Visit 1 of every second cycle, EOT, Visit 1 of every second cycle in FTE, at the EOFT visit (in refractory or relapsed AML patients) and


© 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies. All rights reserved.

Boehringer Ingelheim BI Trial No.: 1315.1 Doc. No.: c02543230-04 28 Apr 2016

Trial Protocol 

during follow-up.

Biochemistry Glucose, sodium, potassium, calcium, inorganic phosphate,

creatinine, AST, ALT, alkaline phosphatase (AP), lactate dehydrogenase (LDH), bilirubin, urea, total protein, albumin,

uric acid

Serum immunoglobulin levels (IgG, IgM, IgA) and direct antiglobulin test have to be measured only every 8 weeks, at

the EOT visit and during follow-up.

Coagulation Activated partial thromboplastin time (aPTT), prothrombin

time (PT), international normalised ratio (INR) where indicated (e.g. treatment with vitamin K antagonists)

Urine pH, glucose, erythrocytes, leukocytes, protein, nitrite will be

analysed by dipstick and reported as semiquantitative measurements. In case of pathological findings, further evaluation should be performed and results documented.

Pregnancy test A serum pregnancy test needs to be obtained at the time

points indicated in the Flow Chart in patients of childbearing

potential.

An additional safety lab will be collected on day 2 of Cycle 1 (i.e., 24 hours after the first administration of BI 836858). Other lab tests to be included: haptoglobin, direct antiglobulin test, bilirubin (direct and indirect) and free hemoglobin. Non pre-existing abnormal laboratory values (CTCAE Grade 3 or higher) will be followed up every 48 hours until these laboratory values are back to at least CTCAE Grade 1.

In case an administration is delayed due to an AE, the patient should visit the site at least once a week for assessment of safety laboratory and AEs. More frequent visits may be appropriate as assessed by the Investigator.

#### 5.2.4 Electrocardiogram

A 12-lead resting ECG will be performed in all patients according to the schedule in the <u>Flow Charts</u>. The ECG will be assessed for pathological results (to be recorded as either concomitant disease or AE) by the Investigator. Additional examinations should be done whenever the Investigator deems necessary.

### 5.2.5 Assessment of other safety parameters

## 5.2.5.1 Vital signs

Vital signs (blood pressure, heart rate and body temperature) will be recorded at every visit during screening, treatment (including the EOT visit) and follow-up. Additional time points for blood pressure and heart rate at the day of administration of BI 836858 are: prior to the start of premedication, prior to the start of BI 836858 infusion, and in 30 ( $\pm$ 10) minute intervals throughout the course of the infusion of BI 836858 and 60 ( $\pm$ 10) minutes after the end of the infusion, thereafter every 4-8 hours until at least 24 hours after start of the infusion. In case of an infusion-related reaction, the Investigator should decide whether to intensify or prolong monitoring of vital signs of the patient.

Beginning with infusion 2, blood pressure and heart rate will be assessed at the same time points as during infusion 1 with the exception that they will not be assessed every 4-8 hours until at least 24 hours after the start of the infusion.

### 5.2.5.2 Physical examination

A physical examination including height, weight and ECOG performance score will be performed at screening and at the time points specified in the Flow Charts. During the physical examination, the patient should be assessed for possible AEs.

## 5.4 APPROPRIATENESS OF MEASUREMENTS

Determination of MTD is based on toxicities graded according to CTCAE (R09-2850). The CTCAE criteria are commonly used in the assessment of AEs in cancer patients. The criteria

Boehringer Ingelheim
BI Trial No.: 1315.1

to be used for evaluation of response ( $\underline{R06-0452}$ ) are well established and scientifically accepted.

Boehringer Ingelheim
BI Trial No.: 1315.1

Boehringer Ingelheim 28 Apr 2016 BI Trial No.: 1315.1

Boehringer Ingelheim
BI Trial No.: 1315.1

Boehringer Ingelheim
BI Trial No.: 1315.1

## 6. INVESTIGATIONAL PLAN

#### 6.1 VISIT SCHEDULE

During the treatment phase, patients with refractory or relapsed AML will receive administration with BI 836858 every 7 days. For AML patients in CR, The first three administrations will be given once every second week on day 1 of Cycles 1, 2 and 3. From the 4<sup>th</sup> administration onwards, patients will receive monthly (every second cycle) infusions of BI 836858 (i.e. 4<sup>th</sup> infusion on Cycle 5 Day 1, 5<sup>th</sup> infusion on Cycle 7 Day 1 ...) for overall up to 12 months of treatment.

Patients are required to be hospitalized under close surveillance with access to intensive care for at least 24 hours after the first administration of BI 836858 to allow close monitoring for infusion-related reactions or other AEs. After good tolerability of the first administration of BI 836858, the Investigator may evaluate the risk for an infusion-related reaction and other AEs in view of relevant co morbidities or AML-related symptoms, and as a result, the patient may receive subsequent infusions in the out-patient setting.

In case a patient misses a visit within one treatment cycle and the patient comes to the clinic between the missed and the next scheduled visit, the delayed visit should be scheduled as soon as possible and documented with the actual date and the reason for the delayed visit. The next visit, should still take place at the time it was originally scheduled in this treatment cycle.

However, in case the day of treatment administration (Visit 1 of a cycle) is delayed, all subsequent visits of a cycle will be recalculated based on the actual date of Visit 1 of the delayed cycle.

## 6.2 DETAILS OF TRIAL PROCEDURES AT SELECTED VISITS

The investigations as outlined in the <u>Flow Charts A</u> and <u>B</u> will be performed at the respective visits as described in detail in the following sections.

## 6.2.1 Screening and run-in period

The screening period (Visit 1), i.e. the phase after informed consent and before the first administration of the trial drug, may be as long as 14 days.

The following parameters and investigations will be obtained and / or performed for <u>both</u> patient populations:

- Informed consent
- Informed consent for pharmacogenetics
- Demographics (sex, birth date, race) and baseline conditions
- Medical history (oncological and relevant non-oncological)
- Review of inclusion and exclusion criteria (patient eligibility)

- Dose assignment (during cohort dose escalation phase only, before the first administration of the trial drug and after informed consent and review of in- and exclusion criteria)
- Safety laboratory (hematology, biochemistry including serum immunoglobulin levels and direct antiglobulin test, coagulation, urine; for details please refer to Section 5.2.3.1)
- Physical examination, height, weight, vital signs and ECOG performance score
- Serum pregnancy test in women of childbearing potential
- 12-lead ECG
- Concomitant therapy
- Bone marrow aspiration for disease assessment (for refractory or relapsed AML patients)

## 6.2.1.1 Re-screening

Sites will be allowed to re-screen patients after 1 week from when they screen failed. If more than 4 weeks have elapsed prior to re-screening, all screening procedures must be repeated.

## 6.2.2 Treatment periods for refractory or relapsed AML patients

6.2.2.1 Visit 1 and Visit 3 – day of BI 836858 administration (administrations 1-8)

On the treatment days, the following parameters and investigations will be obtained and / or performed:

- Review of inclusion and exclusion criteria (patient eligibility), prior to the first administration only
- Safety lab parameters before trial drug administration as specified in <u>Section 5.2.3.1</u>. An additional safety lab will be collected on day 2 of Cycle 1 (i.e., 24 hours after the first administration of BI 836858). Other lab tests to be included: haptoglobin, direct antiglobulin test, bilirubin (direct and indirect) and free hemoglobin. Non pre-existing abnormal laboratory values (CTCAE Grade 3 or higher) will be followed up every 48 hours until these laboratory values are back to at least CTCAE Grade 1.
- Physical examination completed every second cycle beginning with cycle 1. Physical exam may be completed up to 2 days prior to administration and ECOG must be completed on the day of the administration. Height and weight (only at Day 1 of first cycle). If the first administration is completed within 3 days of the screening visit, these examinations do not need to be repeated.
- Vital signs at time points specified in <u>Section 5.2.5.1</u>
- Serum pregnancy test in women of childbearing potential (required at odd-numbered administrations e.g. 1, 3, 5, 7).
- 12-lead ECG (required at Visit 1 of each cycle)
- Adverse events (AEs)

- Changes in concomitant therapies
- Bone marrow aspiration (Required before the 5<sup>th</sup> and 9<sup>th</sup> administration of BI 836858 and at the discretion of the Investigator).

- Administration of BI 836858 after final confirmation of dose tier
- Eligibility for further administration may be performed up to 2 days prior to this visit (at administration 2 and beyond).
- 6.2.2.2 Visit 2 and Visit 4 (± 1 day window allowed beginning in Cycle 3), following administration of BI 836858

In Cycles 1 and 2, visits will occur at Day 4 and Day 11 after the administration. Beginning in Cycle 3 and thereafter, patients will come to the clinic only for infusions and will not be required to complete the visits on Day 4 and Day 11 unless medically indicated. On the Visit 2 and Visit 4 days, the following parameters and investigations will be obtained and / or performed:

- Safety lab parameters before trial drug administration as specified in <u>Section 5.2.3.1</u>
- Vital signs at time points specified in Section 5.2.5.1
- Adverse events (AEs)
- Changes in concomitant therapies

# 6.2.3 End of treatment and follow-up period for refractory or relapsed AML patients

#### 6.2.3.1 EOT visit

This visit includes an evaluation for further treatment. Those patients with clinical benefit after 8 administrations and who are tolerating the infusions well may continue until PD or other criteria for withdrawal are met as noted in Section 3.3.4.1. For those patients who will receive more than 8 administrations, this visit is to be performed 7 days ( $\pm$  2 days) after the 8<sup>th</sup> administration of BI 836858. For those patients who receive <8 administrations, this visit is to be performed 14 days ( $\pm$  2 days) after the last administration of BI 836858.

If the patient concludes the trial within a treatment cycle not at the end of a treatment cycle, the information required to be collected at the EOT visit should be obtained immediately.

The following parameters and investigations will be obtained and /or performed:

- Safety lab parameters and urine analysis as specified in <u>Section 5.2.3.1</u>
- Physical examination, weight
- Vital signs at time points specified in Section 5.2.5.1
- Serum pregnancy test in women of childbearing potential.
- 12-lead ECG
- Adverse events (AEs)
- Changes in concomitant therapies
- Bone marrow aspiration.
- Eligibility for further administration may be performed up to 2 days prior to this visit.
- End of active trial treatment. This will include the reason for conclusion of trial if applicable, premature discontinuation of trial, and date of last administration of the trial drug.

## 6.2.3.2 Further treatment (Visit 1 and Visit 2)

These visits are only for those patients with clinical benefit after 8 administrations and who are tolerating the infusions well. Patients can receive further treatment once the result from the bone marrow assessment from EOT is available. Procedures already done at EOT (i.e., safety lab, pregnancy test) do not need to be repeated at FTE if FTE visit is within 7 days from EOT. The patients will continue to receive weekly infusions until PD or other criteria for withdrawal are met as noted in Section 3.3.4.1.

Prior to each infusion, the following parameters and investigations will be obtained and /or performed:

- Safety lab parameters before trial drug administration as specified in Section 5.2.3.1
- Physical examination every other cycle starting with cycle 5 (may be completed up to 2 days prior) and ECOG performance score.
- Vital signs at time points specified in Section 5.2.5.1
- Serum pregnancy test in women of childbearing potential (required at odd-numbered administrations e.g. 9, 11, 13 etc.)
- Adverse events (AEs)
- Changes in concomitant therapies
- Administration with BI 836858
- Eligibility for further administration may be performed up to 2 days prior to this visit.

Trial Protocol 

#### 6.2.3.3 End of further treatment

This visit is only for those patients who received administrations in further treatment and should be performed 14 days ( $\pm$  2 days) after the last administration of BI 836858.

ECG, bone marrow aspiration, will be performed at EOFT only if the patient has completed at least 2 cycles (e.g. received 4 administrations) since the EOT visit.

The following parameters and investigations will be obtained and /or performed:

- Safety lab parameters and urine analysis as specified in <u>Section 5.2.3.1</u>
- Physical examination including weight (may be completed up to 2 days prior)
- Vital signs at time points specified in <u>Section 5.2.5.1</u>
- Serum pregnancy test in women of childbearing potential
- 12 lead ECG (completed only in patients who receive at least 4 administrations since EOT visit)
- Adverse events (AEs)
- Changes in concomitant therapies
- Bone marrow aspirate (completed only in patients who receive at least 4 administrations since EOT visit)

## 6.2.4 Treatment period for AML patients in CR

## 6.2.4.1 Visit 1– Day 1 of BI 836858 administration (administrations 1-3)

On the treatment days, the following parameters and investigations will be obtained and / or performed:

- Review of inclusion and exclusion criteria (patient eligibility), prior to the first administration only
- Safety lab parameters before trial drug administration as specified in <u>Section 5.2.3.1</u>. An additional safety lab will be collected on day 2 of Cycle 1 (i.e., 24 hours after the first administration of BI 836858). Other lab tests to be included: haptoglobin, direct antiglobulin test, bilirubin (direct and indirect) and free hemoglobin. Non pre-existing abnormal laboratory values (CTCAE Grade 3 or higher) will be followed up every 48 hours until these laboratory values are back to at least CTCAE Grade 1.
- Physical examination and ECOG performance score completed every second cycle
  beginning with cycle 1. Physical exam may be completed up to 2 days prior to
  administration and ECOG must be completed on the day of the administration. Height
  and weight (only at Day 1 of first cycle). If the first administration is completed within 3
  days of the screening visit, these examinations do not need to be repeated.

- Vital signs at time points specified in Section 5.2.5.1
- Serum pregnancy test in women of childbearing potential (required at odd-numbered administrations e.g. 1, 3, 5, 7).
- 12-lead ECG (required at Visit 1 of each cycle)
- Adverse events (AEs)
- Changes in concomitant therapies
- Bone marrow aspiration (at the discretion of the Investigator).
- Peripheral blood for disease assessment. If suspicion of relapse, bone marrow aspiration (or biopsy) for disease assessment is to be performed.
- Administration of BI 836858 after final confirmation of dose tier
- Eligibility for further administration may be performed up to 2 days prior to this visit (at administration 2 and beyond).

#### 6.2.4.2 Further treatment

These visits are only for those patients who have received 3 infusions and are tolerating the infusions well. Patients can receive further treatment every second cycle (i.e., Cycle 5 Day 1, Cycle 7 Day 1, etc.). The patients will continue to receive monthly infusions for overall up to one year of treatment or until PD or other criteria for withdrawal are met (as noted in Section 3.3.4.1).

Prior to each infusion, the following parameters and investigations will be obtained and /or performed:

- Safety lab parameters before trial drug administration as specified in Section 5.2.3.1
- Physical examination every other cycle starting with cycle 5 (may be completed up to 2 days prior)
- Vital signs at time points specified in Section 5.2.5.1
- 12-lead ECG (required at Visit 1 of each cycle)
- Serum pregnancy test in women of childbearing potential (required at odd-numbered administrations e.g. 5, 7, 9 etc.)
- Adverse events (AEs)
- Changes in concomitant therapies
- Peripheral blood for disease assessment. If suspicion of relapse, bone marrow aspiration (or biopsy) for disease assessment is to be performed.
- Administration with BI 836858
- Eligibility for further administration may be performed up to 2 days prior to this visit.

## 6.2.4.3 End of Treatment (EOT) visit

The EOT visit will be performed as soon as possible but no later than one week (7 days) after permanent discontinuation of trial medication for any reason, or when the Investigator decides with the patient to permanently discontinue the trial medication.

If the patient concludes the trial within a treatment cycle not at the end of a treatment cycle, the information required to be collected at the EOT visit should be obtained immediately.

The following parameters and investigations will be obtained and /or performed:

- Safety lab parameters and urine analysis as specified in <u>Section 5.2.3.1</u>
- Physical examination, weight
- Vital signs at time points specified in <u>Section 5.2.5.1</u>
- Serum pregnancy test in women of childbearing potential.
- 12-lead ECG
- Adverse events (AEs)
- Changes in concomitant therapies
- Bone marrow aspiration.
- Peripheral blood for disease assessment. If suspicion of relapse, bone marrow aspiration (or biopsy) for disease assessment is to be performed.
- End of active trial treatment. This will include the reason for conclusion of trial if applicable, premature discontinuation of trial, and date of last administration of the trial drug.
- In case the patient receives further anti-cancer treatment: regimen, drug name and start and stop dates

## 6.2.4.4 End of Residual Effect Period visit (EoR)

The REP is defined in <u>Section 5.2.2.2</u>. The End of REP (EoR) visit should not be performed earlier than 30 days after permanent discontinuation of the trial medication. The information collected at this visit should include all new reportable AEs that occurred after EOT and a follow-up of adverse events ongoing at EOT.

The following parameters and investigations will be obtained and / or performed:

- Date and type of contact
- Vital Signs
- Safety laboratory parameters only if not within normal range at EOT
- 12-lead ECG only if abnormal at EOT and pathological findings were not present at baseline


© 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies. All rights reserved.
- Follow-up of adverse events in case they were not yet recovered at EoT visit
- Documentation of concomitant medications only if indicated for treatment of adverse events
- In case the patient receives further anti-cancer treatment: regimen, drug name and start and stop dates

## **6.2.5** Follow up

Follow up (FU) visits will be performed for <u>both</u> patient populations. These visits will occur after the patient has completed treatment according to protocol or is not eligible for further treatment cycles. These follow-up visits will begin 4 weeks after the last infusion with BI 836858. In patients with AML in CR, follow-up visit 1 (FU1) is the same as EoR. Follow up will end in case the patient is lost to follow-up or in case the Investigator and Sponsor agree not to pursue further follow up visits. Follow up visits should be performed at 4 week intervals or earlier if appropriate as determined by the Investigator.

Follow-up visits should be completed at the investigational site but may be performed by telephone interview in case the patient is unable to visit the Investigator. Follow-up visits should be performed for 6 months after the last infusion with BI 836858. At the last follow-up visit, and end of trial assessment will be performed and documented in the eCRF. For follow-up of patients with adverse events which have not recovered at the last planned follow-up visit please refer to Section 5.2.2.2.

The following will be obtained and / or performed:

- Safety laboratory (hematology, biochemistry including serum immunoglobulin levels and direct antiglobulin test, coagulation, urine; for details please refer to Section 5.2.3.1)
- Physical examination, vital signs.
- AEs since last visit in case they occurred during the observational period (42 days after the last trial drug administration in refractory or relapsed AML patients) or residual effect period (REP, 30 days after the last trial drug administration) or are considered drug-related (see Section 5.2.2.1)
- Concomitant therapy indicated for treatment of an AE
- Follow-up of AEs in case they were not yet recovered at EOT
- Bone marrow aspirate, if indicated
- Treatment with any other anti-leukemia drug (report date of treatment and drug)
- Vital status evaluated at each follow up visit

#### 6.2.6 End of the whole trial

The clinical trial will be analysed and reported after the last patient has completed 4 treatment cycles or stopped treatment prior to completion of cycle 4. In case the trial is ended by the


© 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies. All rights reserved.

Boehringer Ingelheim
28 Apr 2016
BI Trial No.: 1315.1

Sponsor when patients are still being treated with BI 836858 when the final report of the trial is being prepared, the patients will either be included in a follow-up trial or alternatively kept on treatment in this trial. Those patients will then be reported in a revised report and it will be noted in the original report that such a revised report will be written.

28 Apr 2016

Trial Protocol 

# 7. STATISTICAL METHODS AND DETERMINATION OF SAMPLE SIZE

## 7.1 STATISTICAL DESIGN - MODEL

This trial will be performed as an open-label study. The primary objective of the trial is to determine the MTD of BI 836858 for both patient populations separately. To determine the MTD, patients are entered sequentially into escalating dose tiers using the 3+3 design (see Section 3.1). After the MTD has been determined, up to 12 patients for each patient population are additionally entered at this dose level to better characterize the safety of BI 836858.

## 7.2 NULL AND ALTERNATIVE HYPOTHESES

The analyses in this trial are descriptive and exploratory. No formal statistical tests will be performed.

#### 7.3 PLANNED ANALYSES

For the determination of the MTD, only MTD evaluable (i.e. non-replaced patients) will be considered.

For the analysis of secondary all patients in the treated set (i.e. patients treated with at least one dose of BI 836858) will be included in the analysis, including the patients who have been replaced for any reason (see Section 3.3.4.1).

## 7.3.1 Primary analyses

The primary objective for this study is to identify the MTD (for both patient populations separately) and to investigate the safety profile of BI 836858. MTD is defined in Section 3.1, and will be identified by the occurrence of DLT in the dose escalation scheme. In order to identify the MTD, the number of patients with a DLT during the first two cycles at each dose level will be presented. Patients who discontinue during the first two treatment cycles for reasons other than DLT will be excluded from the determination of MTD.

However, for those patients who receive more than two cycles of BI 836858, all AEs that constitute a DLT will be taken into consideration for the purpose of determining the recommended dose for the expansion cohort or the recommended dose for subsequent phase II trial(s).

DLT is defined in <u>Section 5.2.1.1</u>. For the analysis of the tolerability and safety, please refer to <u>Section 7.3.3</u>.

The primary analysis will take place when all patients from the dose escalation and dose expansion cohorts have had a minimum of 4 cycles or have discontinued from the trial prior to reaching end of cycle 4 due to meeting the criteria for withdrawal as outlined in Section 3.3.4.1.

Boehringer Ingelheim 28 Apr 2016 BI Trial No.: 1315.1

In case patients are still being treated at the time of the primary analysis, a revised clinical trial report (CTR) will be created when the last patient has completed his/her last visit, including all primary and secondary analyses.

#### 7.3.2 Secondary analyses

This section outlines the analyses for the secondary defined in <u>Section 5.1.1</u>.

as

## 7.3.2.3 Best overall response

Each patient will be assigned to one of the response categories described in Section 5.1.2.3. Each patient's best overall response will be used as a primary measure. To describe response over time, the proportion of patients in each response category will be tabulated at specified time intervals. The number of patients with objective response (best response of CR, CRi, or PR) will be summarized. Patients will be followed up for assessment of response and progression until they progress, receive any other anti-leukemia therapy, die, or until the trial ends. The observed length of follow-up and the number of patients available for analysis at each time point will determine the period of time covered in tables and figures. Frequency distribution and other descriptive statistical measures will be used to examine these variables.

#### 7.3.2.4 Progression free survival, time to treatment failure

These time-to-event variables will be analyzed with the Kaplan-Meier method.

In case there is no occurrence of death, progression or treatment failure until the last visit of the trial the time will be censored. The percentage of patients who are event free will be displayed at monthly or greater time intervals as appropriate. Details of censoring rules will be provided in the statistical analysis plan.

The cause of death will be summarized, along with whether death was plausible related to disease progression.

## 7.3.3 Safety analyses

Adverse events will be coded using the Medical Dictionary for Regulatory Activities (MedDRA) coding dictionary. Standard BI summary tables and listings will be produced. All adverse events with an onset between start of treatment and end of the residual effect period (REP), a period of 30 days after the last dose of trial medication, will be assigned to the treatment period for evaluation.

All treated patients will be included in the safety analysis. In general, safety analyses will be descriptive in nature and will be based on BI standards. No hypothesis testing is planned.

Statistical analysis and reporting of adverse events will concentrate on treatment-emergent adverse events. To this end, all adverse events occurring between start of treatment and end of the residual effect period will be considered 'treatment-emergent'. The residual effect period is defined as a period of 30 days after the last dose of trial. Adverse events that start before first drug intake and deteriorate under treatment will also be considered as 'treatment-emergent'.

Frequency, severity, and causal relationship of adverse events will be tabulated by system organ class and preferred term after coding according to the current version of the Medical Dictionary for Drug Regulatory Activities (MedDRA).

Laboratory data will be analysed both quantitatively as well as qualitatively. The latter will be done via comparison of laboratory data to their reference ranges. Values outside the reference range as well as values defined as clinically relevant will be highlighted in the listings. Treatment groups will be compared descriptively with regard to distribution parameters as well as with regard to frequency and percentage of patients with abnormal values or clinically relevant abnormal values.

Vital signs, physical examinations, or other safety-relevant data observed at screening, baseline, during the course of the trial and at the end-of-trial evaluation will be assessed with regard to possible changes compared to findings before start of treatment.

## 7.3.4 Interim analyses

The sponsor will continuously monitor safety. The dose escalation design foresees that regular safety evaluations are performed. These evaluations will be un-blinded to dose.

No formal interim analysis of efficacy data is foreseen, although efficacy data when available may be considered as part of the safety evaluations.

28 Apr 2016

As patients with refractory or relapsed AML are known to have low monocyte counts and functional abnormalities of NK cells, both of which are required for the mode of action of BI 836858 (see Section 2.1), detailed evaluations will be performed to ensure a positive benefit-risk assessment in this patient population. If considered unjustifiable, treatment of patients with refractory or relapsed AML may be terminated based on these interim evaluations.

Results of this evaluation of patients with refractory or relapsed AML will be documented and stored. If applicable, the format and the detailed content of the analysis will be defined in the statistical analysis plan.

If considered necessary, a preliminary safety evaluation may also be performed in AML patients in CR. This analysis will have no impact on the further conduct of the trial but can become necessary for internal project purposes. Results of this evaluation will be documented and stored. If applicable the format and the detailed content of such a preliminary analysis will be defined in the statistical analysis plan.

28 Apr 2016

#### 7.4 HANDLING OF MISSING DATA

Every effort will be made to obtain complete information on all AEs, with particular emphasis on potential DLT.

If not stated otherwise, missing data will not be imputed and remain missing. Potential outliers will be reported and analyzed as observed.

The occurrence of missing data should be minimized by follow-up of patients for both disease progression and mortality after end of trial for an individual patient. Both response and progression status for patients who are lost to follow-up or who die before progression has been documented, will be assessed at the end of the trial.

Missing baseline laboratory values will be imputed by respective values from the screening visit.

Trial Protocol 

#### 7.5 RANDOMISATION

This is a non-randomized Phase I trial. All the patients will receive BI 836858.

## 7.6 DETERMINATION OF SAMPLE SIZE

## Patients with refractory or relapsed AML:

Assuming 4 cohorts of 3 patients (i.e. no patients with DLT at given level) and 2 cohorts of 6 patients (i.e. 1 DLT witnessed in first 3 patients so further 3 patients exposed with no DLTs), 24 evaluable patients will be necessary for the dose escalation part.

Together with an assumed number of 12 additional patients for the expansion cohort this leads to an expected sample size of 36 evaluable patients.

## AML patients in CR:

Assuming 1 cohort of 3 patients (i.e. no patients with DLT at given level) and 2 cohorts of 6 patients (i.e. 1 DLT witnessed in first 3 patients so further 3 patients exposed with no DLTs), 15 evaluable patients will be necessary for the dose escalation part in this patient population.

Together with an assumed number of 12 additional patients for the expansion cohort this leads to an expected sample size of 27 evaluable AML patients in CR.

Note that in general, the sample size is induced by the 3+3 design and is subject to different random factors

Doc. No.: c02543230-04  **Trial Protocol** 

#### 8. INFORMED CONSENT, DATA PROTECTION, TRIAL RECORDS

The trial will be carried out in compliance with the protocol, the principles laid down in the Declaration of Helsinki, in accordance with the ICH Harmonised Tripartite Guideline for Good Clinical Practice (GCP) and relevant BI Standard Operating Procedures (SOPs). Standard medical care (prophylactic, diagnostic and therapeutic procedures) remains in the responsibility of the treating physician of the patient.

The Investigator should inform the Sponsor immediately of any urgent safety measures taken to protect the study subjects against any immediate hazard, and also of any serious breaches of the protocol/ICH GCP.

The rights of the Investigator and of the Sponsor with regard to publication of the results of this trial are described in the Investigator contract. As a general rule, no trial results should be published prior to finalisation of the Clinical Trial Report.

#### STUDY APPROVAL, PATIENT INFORMATION, AND INFORMED 8.1 **CONSENT**

This trial will be initiated only after all required legal documentation has been reviewed and approved by the respective Institutional Review Board (IRB) / Independent Ethics Committee (IEC) and competent authority (CA) according to national and international regulations. The same applies for the implementation of changes introduced by amendments.

Prior to patient participation in the trial, written informed consent must be obtained from each patient (or the patient's legally accepted representative) according to ICH GCP and to the regulatory and legal requirements of the participating country. Each signature must be personally dated by each signatory and the informed consent and any additional patientinformation form retained by the Investigator as part of the trial records. A signed copy of the informed consent and any additional patient information must be given to each patient or the patient's legally accepted representative.

The patient must be informed that his/her personal trial-related data will be used by Boehringer Ingelheim in accordance with the local data protection law. The level of disclosure must also be explained to the patient.

The patient must be informed that his / her medical records may be examined by authorized CML/Clinical Research Associate (CRA) or Clinical Quality Assurance auditors appointed by Boehringer Ingelheim, by appropriate IEC members, and by inspectors from regulatory authorities.

#### 8.2 DATA QUALITY ASSURANCE

The trial will be conducted in compliance with the protocol, the principles laid down in the Declaration of Helsinki (please, refer to Section 8), local law and according to the principles of GCP and the company SOPs. To inform all Investigators about the trial drugs and the


© 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies. All rights reserved.

Trial Protocol 

procedures of the trial, either an Investigator meeting will be performed prior to start of the trial, or each Investigator will be visited individually by the Clinical Monitor and the CRA. Each Investigator will receive an ISF with all information relevant for the performance of the trial. Investigators will be visited at regular intervals for on-site monitoring by a Boehringer Ingelheim employee or a CRA authorised by BI. At these occasions, source data verification (SDV) will be performed and a check will be done whether the eCRFs are kept current. The information in the eCRF and information in source documents will be cross-checked as described in Section 8.3.1.

The data management procedures to ensure the quality of the data are described in detail in the trial data management and analysis plan (TDMAP) available in the Clinical Trial Master File (CTMF). Coding of the data obtained will be done by using the medical dictionary for regulatory activities (MedDRA) and the WHO dictionary for concomitant medication. Data quality review meetings will be performed at regular intervals to evaluate the quality of the data collected. Discrepancies in data will be queried.

A quality assurance audit/inspection of this trial may be conducted by the Sponsor or Sponsor's designees or by IRBs/IECs or by regulatory authorities. The quality assurance auditor will have access to all medical records, the Investigator's trial-related files and correspondence, and the informed consent documentation of this clinical trial.

## 8.3 RECORDS

Case Report Forms (CRFs) for individual patients will be provided by the Sponsor via remote data capture. For drug accountability, refer to Section 4.1.8.

## **8.3.1** Source documents

Source documents provide evidence for the existence of the patient and substantiate the integrity of the data collected. Source documents are filed at the Investigator's site.

Data entered in the eCRFs that are transcribed from source documents must be consistent with the source documents or the discrepancies must be explained. The Investigator may need to request previous medical records or transfer records, depending on the trial; also current medical records must be available.

For eCRFs all data must be derived from source documents.

#### 8.3.2 Direct access to source data and documents

The Investigator / institution will permit trial-related monitoring, audits, IRB / IEC review and regulatory inspection, providing direct access to all related source data / documents. CRFs/eCRFs and all source documents, including progress notes and copies of laboratory and medical test results must be available at all times for review by the Sponsor's clinical trial monitor, auditor and inspection by health authorities (e.g. FDA). The CRA / on site monitor and auditor may review all CRFs/eCRFs, and written informed consents. The accuracy of the data will be verified by reviewing the documents described in Section 8.3.1.

#### 8.4 LISTEDNESS AND EXPEDITED REPORTING OF ADVERSE EVENTS

#### 8.4.1 Listedness

To fulfil the regulatory requirements for expedited safety reporting, the Sponsor evaluates whether a particular adverse event is "listed", i.e. is a known side effect of the drug or not. Therefore a unique reference document for the evaluation of listedness needs to be provided. For BI 836858 this is the current version of the IB (c02324887-03). The current versions of these reference documents are provided in the ISF.

## 8.4.2 Expedited reporting to health authorities and IECs/IRBs

Expedited reporting of SAEs, e.g. suspected unexpected serious adverse reactions (SUSARs) to health authorities and IECs/IRBs, will be done according to local regulatory requirements. Further details regarding this reporting procedure are provided in the ISF.

## 8.5 STATEMENT OF CONFIDENTIALITY

Individual patient medical information obtained as a result of this trial is considered confidential and disclosure to third parties is prohibited with the exceptions noted below. Patient confidentiality will be ensured by using patient identification code numbers.

Treatment data may be given to the patient's personal physician or to other appropriate medical personnel responsible for the patient's welfare. Data generated as a result of the trial need to be available for inspection on request by the participating physicians, the Sponsor's representatives, by the IEC and the regulatory authority.

## 9. **REFERENCES**

#### 9.1 PUBLISHED REFERENCES

- R01-0028 Simon R, Freidlin B, Rubinstein L, Arbuck SG, Collins J, Christian MC. Accelerated titration designs for phase I clinical trials in oncology. J Natl Cancer Inst. 1997. 89(15): 1138–1147.
- R01-0787 Oken, M.M., Creech, R.H., Tormey, D.C., Horton, J., Davis, T.E., McFadden, E.T., Carbone, P.P.: Toxicity And Response Criteria Of The Eastern Cooperative Oncology Group. Am J Clin Oncol 5:649-655, 1982
- R01-1267 Caron PC, Jurcic JG, Scott AM, Finn RD, Divgi CR, Graham MC, et.al. A phase 1B trial of humanized monoclonal antibody M195 (anti-CD33) in myeloid leukemia: specific targeting without immunogenicity. Blood. 1994. 83(7): 1760-1768.
- R04-0569 Kang SH, Ahn CW. An investigation of the traditional algorithm-based designs for phase 1 cancer clinical trials. Drug Inf J. 2002. 36: 865–873.
- R06-0452 Cheson BD, Bennett JM, Kopecky KJ, Buchner T, Willman CL, Estey EH, et.al. Revised recommendations of the International Working Group for Diagnosis, Standardization of Response Criteria, Treatment Outcomes, and Reporting Standards for Therapeutic Trials in Acute Myeloid Leukemia. J Clin Oncol. 2003. 21(24): 4642-4649.
- R07-2767 Stone RM, O'Donnell MR, Sekeres MA. Acute myeloid leukemia. Hematology. 2004: 98–117.
- R07-2768 Estey E, Doehner H. Acute myeloid leukaemia. Lancet. 2006. 368: 1894-1907.
- R07-2769 NCCN Clinical Practice Guidelines in Oncology: acute myeloid leukemia (V.1.2006). www.nccn.org; National Comprehensive Cancer Network 2005.
- R07-2770 Froehling S, Schlenk RF, Kayser S, Morhardt M, Benner A, Doehner K, et.al. Cytogenetics and age are major determinants of outcome in intensively treated acute myeloid leukemia patients older than 60 years: results from AMLSG trial AML HD98-B. Blood. 2006. 108 (10): 3280–3288.
- R07-2771 Burnett AK, Milligan D, Prentice AG, Goldstone AH, McMullin MF, Hills RK, et.al. A comparison of low-dose cytarabine and hydroxyurea with or without all-trans retinoic acid for acute myeloid leukemia and high-risk myelodysplastic syndrome in patients not considered fit for intensive treatment. Cancer. 2007. 109(6): 1114–1124.
- Estey E. Acute myeloid leukemia and myelodysplastic syndromes in older patients. J Clin Oncol. 2007. 25(14): 1908–1915.

| R07-2773 | Menzin J, Lang K, Earle CC, Kerney D, Mallick R. The outcomes and costs of acute myeloid leukemia among the elderly. Arch Intern Med. 2002. 162: 1597–1603. |
|---|---|
| R07-2774 | Mrozek K, Bloomfield CD. Chromosome aberrations, gene mutations and expression changes, and prognosis in adult acute myeloid leukemia. Hematology. 2006:169–177. |
| R07-2854 | Becker C, Ali HA, Krahl R, Poenisch W, Wedding U, Fiedler, F, et.al. High complete remission rate in patients with acute myeloid leukemia (AML) above the age of 60 years: a report of the AML97#38 study of the East German Hematology and Oncology Study Group. Blood. 2004. 104(11): Abstr 880. |
| R09-2850 | Common terminology criteria for adverse events (CTCAE) version 4.0 (publish date: May 28, 2009). U.S.Department of Health and Human Services, National Institutes of Health, National Cancer Institute (2009). |
| R10-2947 | Dohner H, et.al. Diagnosis and management of acute myeloid leukemia in adults: recommendations from an international expert panel, on behalf of the European LeukemiaNet. Blood, 21 January 2010, Volume 115, Number 3. |
| R10-4428 | Chung CH. Managing premedications and the risk for reactions to infusional monoclonal antibody therapy. Oncologist. 2008. 13: 725-732. |
| R10-4517 | Coiffier B, Altman A, Pui CH, Younes A, Cairo MS. Guidelines for the management of pediatric and adult tumor lysis syndrome: an evidence-based review. J Clin Oncol. 2008. 26(16): 2767-2778. |
| R10-6267 | Wang DD, Zhang S, Zhao H, Men AY, Parivar K. Fixed dosing versus body size-based dosing of monoclonal antibodies in adult clinical trials. J Clin Pharmacol. 2009. 49: 1012-1024. |
| R11-1467 | Crocker PR, Zhang J. New I-type lectins of the CD33-related Siglec subgroup identified through genomics. Biochem Soc Symp. 2002. 69: 83-84.R11-1468 |
| R11-1468 | Scheinberg DA, Tanimoto M, McKenzie S, Strife A, Old LJ, Clarkson BD. Monoclonal Antibody M195: A Diagnostic Marker for Acute Myelogenous Leukemia. Leukemia. 1989. 3: 440-445. |
| R11-1469 | Hauswirth AW, Florian S, Printz D, Sotlar K, Krauth MT, Fritsch G, et.al. Expression of the target receptor CD33 in CD43+/CD38-/CD123+ AML stem cells. Eur J Clin Invest. 2007. 37: 73-82. |
| R11-1470 | Plesa C, Chelghoum Y, Plesa A, Elhamri M, Tidaud I, Michallet M, et.al.<br>Prognostic Value of Immunophenotyping in Elderly Patients with Acute |

Myeloid Leukemia. Cancer. 2007. 112(3): 572-580.

- R11-1471 Raza A, Jurcic JG, Roboz GJ, Maris M, Stephenson JJ, Wood BL, et.al. Complete remission observed in acute myeloid leukaemia following prolonged exposure to lintuzumab: a phase I trial. Leukemia & Lymphoma. 2009: 1-9.
- R11-1472 Lapusan S, Vidriales MB, Thomas X, de Botton S, Vekhoff A, Tang R, Dumontet C, et.al. Phase I studies of AVE9633, an anti-CD33 antibody-maytansinoid conjugate, in adult patients with relapsed/refractory acute myeloid leukemia. Invest New Drugs. 2011 Apr 26.
- R11-1473 Taussig DC, Pearce DJ, Simpson C, Rohatiner AZ, Lister TA, Kelly G, et.al. Hematopoietic stem cells express multiple myeloid markers: implications for the origin and targeted therapy of acute myeloid leukemia. Blood. 2005. 106: 4086-4092.
- R11-1474 Caron PC, Dumont L, Scheinberg DA. Supersaturating Infusional Humanized Anti-CD33 Monoclonal Antibody HuM195 in Myelogenous Leukemia. Clinical Cancer Research. 1998. 4: 1421-1428.
- R11-1481 Raza A, Jurcic JG, Roboz GJ, Maris M, Stephenson JJ, Wood BL, et.al. Complete remissions observed in acute myeloid leukemia following prolonged exposure to lintuzumab: a phase 1 trial. Leukemia & Lymphoma. 2009 Aug. 50(8): 1336-1344.
- Webber BA, Cushing MM, Li S. Prognostic significance of flow cytometric immunophenotyping in acute myeloid leukemia. Int J Clin Exp Pathol. 2008. 1(2): 124-133.
- R11-4256 Caron PC, Co MS, Bull MK, Avdalovic NM, Queen C, Scheinberg DA. Biological and immunological features of humanized M195 (anti-CD33) monoclonal antibodies. Cancer Res. 1992. 52: 6761-6767.
- R11-4695 Jurcic, JG, et.al. Molecular Remission Induction with Retinoic Acid and Anti-CD33 Monoclonal Antibody HuM195 in Acute Promyelocytic Leukemia. Clin can res. February 2000. Vol. 6, 372–380.
- R15-6192 Stringaris K, Sekine T, Khoder A, Alsuliman A, Razzaghi B, Sargeant R, Pavlu J, Brisley G, Lavallade H de, Sarvaria A, Marin D, Mielke S, Apperley JF, Shpall EJ, Rezvani K. Leukemia-induced phenotypic and functional defects in natural killer cells predict failure to achieve remission in acute myeloid leukemia. Haematologica. 2014. 99 (5), 836 847.

## 9.2 UNPUBLISHED REFERENCES

U11-2766-01 Investigator's Brochure: BI 836858 (Version 1.0). 09 December

2011.

c02324887-03 Investigator's Brochure: BI 836858 (Version 5.0). 14 Aug 2015.

28 Apr 2016

## 10. APPENDICES

#### 10.1 PUBLICATION POLICIES

Boehringer Ingelheim is as much as possible dedicated to support process of free exchange of relevant scientific information. Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the Investigator and of the Sponsor with regard to publication of the results of this trial are described in the Investigator contract. As a general rule, no trial results should be published prior to finalisation of the Clinical Trial Report (CTR).

The present trial will be published in a clinical trial registry indicating the trial dates and indication as well as the number of sites and location.

## 10.2 EASTERN COOPERATIVE ONCOLOGY GROUP (ECOG) PERFORMANCE STATUS

## **ECOG PERFORMANCE STATUS (R01-0787)**

| Grade | ECOG |
|---|---|
| 0 | Fully active, able to carry on all pre-disease performance without restriction |
| 1 | Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work |
| 2 | Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours |
| 3 | Capable of only limited self-care, confined to bed or chair more than 50% of waking hours |
| 4 | Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair |
| 5 | Dead |

## 10.3 CLINICAL EVALUATION OF LIVER DISEASE

#### 10.3.1 Introduction

Alterations of liver laboratory parameters, as described in <u>Section 5.2.2.1</u> (Protocol-Specified Significant Events), are to be further evaluated using the following procedures:

#### 10.3.2 Procedures

Repeat the following lab tests: ALT, AST, and bilirubin (total and direct) - within 48 to 72 hours. If ALT and/or AST >3-fold ULN combined with an elevation of total bilirubin >2-fold ULN are confirmed, results of the laboratory parameters described below must be made available to the Investigator and to BI as soon as possible.

#### In addition,

- obtain a detailed history of current symptoms and concurrent diagnoses and medical history according to the "Drug Induced Liver Injury (DILI) checklist" provided in the ISF
- obtain history of concomitant drug use (including non-prescription medications, herbal and dietary supplement preparations), alcohol use, recreational drug use, and special diets according to the "DILI checklist" provided in the ISF;
- obtain a history of exposure to environmental chemical agents (consider home and work place exposure) according to the "DILI checklist" provided in the ISF; and report these via the CRF.

## Clinical chemistry

Alkaline phosphatase, albumin, PT or INR, CK, CK-MB, coeruloplasmin, α-1 antitrypsin, transferin, amylase, lipase, fasting glucose, cholesterol, triglycerides

#### Serology

Hepatitis A (Anti-IgM, Anti-IgG), Hepatitis B (HbsAg, Anti-HBs, DNA), Hepatitis C (Anti-HCV, RNA if Anti-HCV positive), Hepatitis D (Anti-IgM, Anti-IgG), Hepatitis E (Anti-HEV, Anti-HEV IgM, RNA if Anti-HEV IgM positive), Anti-Smooth Muscle antibody (titer), Anti-nuclear antibody (titer), Anti-LKM (liver-kidney microsomes) antibody, Antimitochondrial antibody

Hormones, tumor marker TSH

## Haematology

Thrombocytes, eosinophils

• Provide abdominal ultrasound to rule out biliary tract, pancreatic or intrahepatic pathology, e.g. bile duct stones or neoplasm.

Boehringer Ingelheim 28 Apr 2016 BI Trial No.: 1315.1

• Initiate close observation of subjects by repeat testing of ALT, AST, and total bilirubin (with fractionation by total and direct) at least weekly until the laboratory ALT and/or AST abnormalities stabilize or return to normal, then according to the protocol. Depending on further laboratory changes, additional parameters identified e.g. by reflex testing will be followed up based on medical judgment and Good Clinical Practice (GCP).

## 11. DESCRIPTION OF GLOBAL AMENDMENTS

| Number of global amendment | 01 |
|---|---|
| Date of CTP revision | 13 April 2012 |
| EudraCT number | N/A |
| BI Trial number | 1315.1 |
| BI Investigational Product(s) | BI 836858 |
| Title of protocol | A Phase I, open, cohort dose escalation trial with BI 836858 in patients with refractory or relapsed acute myeloid leukemia |
| To be implemented only after approval of the IRB/IEC/Competent Authorities | |
| To be implemented immediately in order to eliminate hazard — IRB / IEC / Competent Authority to be notified of change with request for | |
| approval | |
| Can be implemented without IRB/IEC/ Competent Authority approval as changes involve logistical or administrative aspects only | |
| Section to be changed | Title page |
| Description of change | Change of TCM and contact information; <u>Status</u> : "Final Protocol" has been removed and "Revised Protocol (based on Global Amendment 01)" has been added <u>Version and Date</u> : Version 1.0 has been replaced with Version 2.0 |
| Rationale for change | Clarification and update |
| Section to be changed | Section 3.3.3 Exclusion Criteria |
| Description of change | The following exclusion criterion has been added: |
| | Patients who are candidates for allogeneic stem |
| | cell transplantation. |
| Rationale for change | Clarification that all eligible patients should have |

| Number of global amendment | 01 |
|---|---|
| | received all standard therapies available for AML, |
| | before participating in a first in human trial |
| Section to be changed | Section 4.1.3 Selection of doses in the trial and |
| _ | Table 4.1.3: 1 Entry of patients into trial, by |
| | cohort |
| Description of change | Section 4.1.3: Clarification of the cohort dose |
| | escalation phase for enrolment of patients into the |
| | first dose cohort of 10 mg |
| | <u>Table 4.1.3: 1</u> : Addition of footnote for |
| | clarification of cohort dose escalation phase for |
| | enrolment of patients into the first dose cohort of |
| | 10 mg |
| Rationale for change | Clarification |

Boehringer Ingelheim 28 Apr 2016

BI Trial No.: 1315.1

| Number of global amendment | 02 |
|---|---|
| Date of CTP revision | 14 Jun 2013 |
| EudraCT number | N/A |
| BI Trial number | 1315.1 |
| BI Investigational Product(s) | BI 836858 |
| Title of protocol | A Phase I, open, cohort dose escalation trial with BI |
| Title of protocol | 836858 in patients with refractory or relapsed acute |
| | myeloid leukemia |
| To be implemented only after | |
| approval of the | |
| IRB/IEC/Competent | |
| Authorities | |
| To be implemented | |
| immediately in order to | |
| eliminate hazard – | |
| IRB / IEC / Competent | |
| Authority to be notified of | |
| change with request for | |
| approval | |
| Can be implemented without | |
| IRB/IEC/ Competent | |
| Authority approval as changes | |
| involve logistical or | |
| administrative aspects only | |
| | Tr: d |
| Section to be changed | Title page |
| Description of change | Status: "Revised Protocol (based on Global |
| | Amendment 01)" has been updated to be "Revised |
| | Protocol (based on Global Amendments 01 and 02)" |
| | Version and Date: Version 2.0 has been replaced |
| D. C. L. C. L. | with Version 3.0 |
| Rationale for change | Clarification and update |
| Section to be changed | Protocol Synopsis |
| Description of change | Objective: "refractory or relapsed" has been added |
| | Mode of admin: the time period of the infusion "over 3 hours" was deleted |
| | <u>Duration of treatment</u> : Language has been updated from "Those patients with partial response (PR) or |
| | complete response (CR) after 8 administrations and |
| | who are tolerating the infusions may continue until progressive disease (PD)" to read " <i>Those patients</i> |
| | with clinical benefit as defined by International |
| | Working Group (IWG) objective response (partial |

| Number of global amendment | 02 |
|---|---|
| Number of global amenument | remission (PR) or complete remission (CR) or |
| | complete remission with incomplete blood recovery |
| | (CRi)) or subjective response (in the absence of |
| | objective response) after 8 administrations and who |
| | are tolerating the infusions may continue until |
| | progressive disease (PD)." |
| | <u>Criteria for safety</u> : The following parameters have |
| | been added: "vital signs, ECG, physical |
| | examination and" |
| Rationale for change | Clarification and update |
| Section to be changed | Flow Chart |
| Description of change | <u>Trial Period</u> : "Demographics" has been updated to |
| | "Demographics and baseline conditions", "Adverse |
| | events" has been marked to be collected at |
| | screening, "Pharmacokinetics" and "Anti-drug |
| | antibodies" have been marked to be collected at |
| | further treatment visits, and "Vital Status" has been |
| | added. |
| | Footnotes: EOT footnote replaced "CR" with "CRi |
| | or CR" |
| | ** section has replaced "CR" with "CRi or CR" |
| | Footnote 3 has removed "footnote 1" and replaced with "footnote 2" |
| | Footnote 4 wording has been added: "An additional |
| | safety lab will be collected on day 2 (i.e., 24 hours |
| | after the first administration of BI 836858). Other |
| | lab tests to be included: haptoglobin, direct Coombs |
| | test, and bilirubin (direct and indirect)". |
| | Footnote 10 has been updated to: Bone marrow |
| | aspirate to assess efficacy before 5 <sup>th</sup> and 9 <sup>th</sup> |
| | administrations "(i.e., BM performed on Day 1 (+/- |
| | 1) of cycles 3 and 5 and treatment started on day 1 |
| | (up to $+3$ ) of cycles 3 and 5)" |
| | Footnote 14 has removed "Cycle 1 Day 9, Cycle 2 |
| | Day 2, and Cycle 2 Day 9 in addition to those" and |
| | been updated to "Sampling at the time points |
| | specified in Tables 1 and 2. As noted in Tables 1 |
| | and 2 PK sampling timepoints specify visits on |
| | Cycles 1 and 2 Days 1, 2, 4, 8, 9 and 11 and EOT |
| | and on Cycle $\geq$ 3 Days 1 and 8 and EOT/EOFT as |
| | noted in the Flow Chart. |
| | Footnote 17 has been updated to "After the 8th |
| | infusion, at the end of treatment visit, patients will |
| | be evaluated to determine if they have clinical |

| Number of global amondment | 02 |
|---|---|
| Number of global amendment | |
| | benefit, as defined by IWG objective response (PR, CRi or CR) or subjective response (in the absence of objective response) and are tolerating the infusions well and who would like to continue to receive infusions until PD or other criteria for withdrawal are met as noted in Section 3.3.4.1. For each infusion past the 8th administration, patients will continue to be assessed after each cycle for clinical benefit (objective or subjective response), and that they are tolerating the infusions well and would like to continue until PD or other criteria for withdrawal are met as noted in Section 3.3.4.1." |
| Rationale for change | Clarification and update. |
| | For footnote 4, an additional safety lab was added on day 2, 24 hours after the first administration of BI 836858. The aim is to observe elevated laboratory values earlier and, with additional parameters (e.g. liver enzymes) to better understand the cause of the laboratory values. Non pre-existing abnormal laboratory values (CTCAE Grade 3 or higher) will be followed up every 48 hours until these laboratory values are back to at least CTCAE Grade 1. |
| Section to be changed | Table 1 and Table 2 |
| Description of change | Blood sampling timepoints have been updated in both tables. For Table 2, additional blood sampling timepoints have been added for cycles≥3 |
| Rationale for change | Update |

| Number of global amendment | 02 |
|---|---|
| g | The schedule to investigate cytokine levels at |
| | specific timepoints was adapted following the FDA |
| | guidance (Draft Guidance for Industry |
| | Immunogenicity Assessment for Therapeutic |
| | Protein Products). |
| Section to be changed | Abbreviations |
| Description of change | "ASCT Allogeneic stem cell transplantation" was |
| | added. |
| | In CRi abbreviation, "marrow" was removed and |
| | "blood" was added. |
| | "NK Natural Killer (cells)" was added. |
| Rationale for change | Clarification and update |
| Section to be changed | Section 1.1 Medical Background |
| Description of change | "Objective response was defined as either CR, CRi |
| | or PR" was added |
| Rationale for change | Clarification and update |
| Section to be changed | Section 2.2 Trial Objectives |
| Description of change | Section was revised to read as follows: The primary |
| | objective of this trial is to determine the maximum |
| | tolerated dose (MTD) of BI 836858. BI 836858 is a |
| | new biological entity (NBE) and the MTD may not |
| | be reached. Even if no MTD is reached the highest |
| | dose of BI 836858 that may be tested is 800 mg. To learn more about the safety and preliminary efficacy |
| | there will be an expansion cohort either at the MTD |
| | or 800mg. "the highest tested dose (e.g. 320 mg)." |
| Rationale for change | Clarification and Update |
| Section to be changed | Sections Flow Chart- EOT footnote, 2.2, 3.3.3, |
| Section to be changed | 3.3.4.1, 5.5.1, 5.5.2.1, 5.5.3.2, 5.6, 5.6.2, 5.6.3, |
| | 6.2.2.2, 6.2.3.1, 7.3, 7.3.2.4, 10.3 |
| Description of change | Grammatical and spelling updates |
| Rationale for change | Grammatical and spelling updates |
| Section to be changed | Section 3.1 Overall Trial Design and Plan |
| Description of change | Text was revised and dose levels were modified as |
| 2 escription of change | follows: |
| | "The dose is planned to be escalated in cohorts at |
| | pre-defined dose levels based on a multiplication |
| | factor of 2. 3 in the low dose range, and a factor of |
| | approximately 2 at doses higher than 90 mg. The |
| | dose levels are 10 mg, 20 mg, 40 mg, 80 mg, 160 |
| | mg, and 320 mg <del>10 mg, 30 mg, 90 mg, 200 mg, 400</del> |
| | mg, and 800 mg as outlined in Section 4.1.3. |
| | However, Intermediate dose levels and levels |
| | higher than 320 mg may be investigated if agreed |

Boehringer Ingelheim 28 Apr 2016

BI Trial No.: 1315.1 Doc. No.: c02543230-04 Trial Protocol 

| Number of global amendment | 02 |
|---|---|
| 9 | upon between Investigator and Sponsor." |
| | "In case no MTD is reached up to the highest planned dose (e.g., 320 mg), of 800 mg, 12 additional patients will be treated with once weekly highest test dose (i.e., 320 mg) 800 mg of BI 836858." |
| | Clarification of treatment in the dose escalation phase of the trial as follows: "During the dose escalation phase, each patient will receive up to 2 repeated treatment cycles. In patients who show clinical benefit as defined by IWG objective response (CR, CRi, PR), or subjective response (in the absence of objective response) as defined by the Investigator after 2 cycles, the number of cycles on the same dose level may be increased to 4 (8 administrations) upon agreement between Investigator and Sponsor. This includes Cycle three (administration of BI 836858 on Days 29 and 36) and cycle four (administration of BI 836858 on Days 43 and 50). Continuation of treatment will be discussed between Investigators and Sponsor at each cycle." |
| | Text has been revised as follows: Patients who show "clinical benefit", (CR, CRi, PR, or subjective response) elinical benefit as defined by the Investigator after 4 cycles "(each cycle individually evaluated))," and who are tolerating the infusions well may continue to receive additional cycles upon agreement between Investigator and Sponsor until the patient meets any of the criteria for withdrawal as outlined in Section 3.3.4.1." |
| Rationale for change | Clarification and Update and Safety. To mitigate the risk of dose dependent side effects, all dose levels will be based on a multiplication factor of two (x2) and the doses pre-defined i.e. 10, 20, 40, 80, 160 and 320 mg of BI 836858. |

| Number of global amendment | 02 |
|---|---|
| Section to be changed | Section 3.2 DISCUSSION OF TRIAL DESIGN, |
| | INCLUDING THE CHOICE OF CONTROL |
| | GROUP |
| Description of change | The text was revised as follows: |
| | In case no MTD is reached up to the highest |
| | planned dose (e.g., 320 mg), of 800mg, 12 |
| | additional patients will be treated with once weekly |
| | of the highest tested dose (e.g., 320 mg) 800 mg of |
| | BI 836858. |
| | "And pharmacologic/pharmacodynamic" has been |
| D 4: 1 C 1 | removed from this section. |
| Rationale for change | Clarification and Update |
| Section to be changed | Section 3.3 Selection of trial population |
| Description of change | "About" was added to target of 10 patients. Clarification |
| Rationale for change | |
| Section to be changed | Section 3.3.2 Inclusion Criteria |
| Description of change | Inclusion criteria #2 added "per central laboratory assessment at the Ohio State University". |
| | Inclusion criteria #3 added "See Section 10.2". |
| | Inclusion criteria #4 removed ">" and replaced with |
| | ">". |
| Rationale for change | Clarification |
| Section to be changed | Section 3.3.3 Exclusion Criteria |
| Description of change | Exclusion criterion #2 – text was revised: "Patients |
| | with >30,000 leukocytes/μl in the peripheral blood |
| | was changed to "Patients with >5,000 leukocytes/μl |
| | in the peripheral blood". |
| | Exclusion criterion #3- text was removed and |
| | updated for clarification: "Anti-leukemia therapy |
| | within two weeks before first treatment with BI |
| | 836858; however, parallel treatment with |
| | Hydroxyurea is allowed. (Hydroxyurea may be |
| | given until 48 hours before the first treatment with BI 836858) (See Section 4.2.2.1)" |
| | <del>B1 030030)</del> (See <u>Section 4.2.2.1</u> ) |
| | Exclusion criterion #13 has removed "the evaluation |
| | of efficacy or safety of the trial drug and reads as |
| | follows: "Concomitant intercurrent illness, or any |
| | condition which in the opinion of the Investigator, |
| | would compromise safe participation in the study, |
| | e.g. active severe infection, unstable angina |
| | pectoris, new onset of exacerbation of a cardiac |
| | arrhythmia" |

| Number of global amendment | 02 |
|---|---|
| Rationale for change | Clarification, update and safety. |
| | To control the WBC, a treatment with hydroxyurea |
| | is allowed (as noted in Exclusion #3). The parallel |
| | use of hydroxyurea may allow patients with a |
| | proliferative disease to remain on study. This may |
| | also reduce the number of early study withdrawals, |
| | especially in the lower dose cohorts, as disease |
| | progression may be controlled. |
| Section to be changed | Section 3.3.4.1 Removal of individual patients |
| Description of change | "4 administrations (1 cycle)" has been replaced by |
| | "4 administrations (2 cycles)". |
| Rationale for change | Clarification and correction |
| Section to be changed | Section 4.1 TREATMENTS TO BE ADMINISTERED |
| Description of change | Text was revised to read as follows: BI 836858 will |
| | be administered as an as a rate-controlled |
| | intravenous infusion. |
| | Text was deleted for clarification: (Volume: 250 |
| | mL) <del>, Rate: see Table 4.1.1:1 below)</del> |
| Rationale for change | Posology was revised - update |
| Section to be changed | Section 4.1.1 Identity of BI investigational product |
| | and comparator product |
| Description of change | Posology was revised from "Infusion over 3 hours" |
| | to "Rate controlled infusion". Table 4.1.1: 1 was removed and text was added as |
| | explanation for infusion rate as follows: |
| | "The first and second infusion will be started at a |
| | rate of 10 mL/h. The infusion rate should be |
| | increased every 30 (+/-10) minutes by 10 mL/h to a |
| | maximum of 80 mL/h as long as tolerated by the |
| | patient. If considered safe by the Investigator, the |
| | stepwise increase of infusion rate during the third |
| | and subsequent infusions may be faster or steps may |
| | be omitted, but the maximum infusion rate must not |
| | exceed 120 mL/h. If symptoms of an infusion-related |
| | reaction occur, the infusion should be temporarily |
| | stopped. Upon recovery, it should be infused at 50% |
| | of the rate at which the reaction occurred and |
| | should not be dose escalated from this dose for at |
| | least 30 minutes. Lower rates may be selected if |
| | clinically indicated. Depending on the time of |
| | occurrence and the severity of the reaction, the |
| | investigator may consider administering additional |

| Number of global amendment | 02 |
|---|---|
| | supportive medication, e.g. corticosteroids. A stepwise re-increase of the infusion rate to a maximum of 80 mL/h is possible. For medical reasons, in case a patient experiences an adverse event during the infusion, the duration of the infusion may be expanded until the use-by date and use-by time indicated on the label is reached. The actual duration of the infusions and the infusion steps need to be documented in the eCRF including actual start and end time, actual time points for interruption and restart of the infusion and the actual infusion rates." |
| Rationale for change | Clarification and Update. The stepwise increase of the infusion rate of BI 836858 was adapted and an upper limit of 80ml/hr is defined in the protocol amendment. However, some flexibility is given in case the first four administrations of BI 836858 are well tolerated. |
| Section to be changed | Section 4.1.3 Selection of doses in the trial |
| Description of change | Text was modified as follows: "BI 836858 will be administered as a rate-controlled; intravenous infusion as noted in Table 4.1.1: 1 over 3 hours every 7 days." The text referring to dose levels was modified: "The dose is planned to be escalated in cohorts at predefined dose levels based on a multiplication factor of 2. 3 in the low dose range, and a factor of approximately 2 at doses higher than 90 mg. The dose levels are 10 mg, 30 mg, 90 mg, 200 mg, 400 mg, and 800 mg. However, The dose levels are 10 mg, 20 mg, 40 mg, 80 mg, 160 mg, and 320 mg. Intermediate dose levels and dose levels higher than 320 mg may be investigated if agreed upon between Investigator and Sponsor. Clarification that enrolment into the next highest dose cohort has been corrected from "14 days" to "28 days". Text was modified: In case no MTD is reached up to the highest planned tested dose (e.g. 320 mg), of 800 mg, 12 additional patients will be treated with |

| Number of global amendment | 02 |
|---|---|
| | once weekly with the highest tested dose (e.g. 320 mg) 800 mg of BI 836858 in the expansion cohort. |
| Rationale for change | Clarification and update To mitigate the risk of dose dependent site effects, all dose levels will be based on a multiplication factor of two (x2) and the doses pre-defined i.e. 10, 20, 40, 80, 160 and 320 mg of BI 836858. |
| Section to be changed | Section 4.1.4 Drug assignment and administration of doses for each patient |
| Description of change | Updated glucocorticoid i.v., equivalent to prednisolone dose from "50mg" to "100mg" Language updated to read as follows: "If BI 836858 has been well tolerated without signs of infusion-related reactions in the first administration, glucocorticoid premedication may be reduced to a dose equivalent to 25 50 mg prednisolone for the second through fourth administrations, and in case this is well tolerated reduce the steroids with the 5th infusion (25 mg with 5th and 0 mg with the 6th infusion.) However, in case an administration of BI 836858 was not well tolerated the premedication with prednisolone can be re-escalated up to 100 mg." |
| Rationale for change | Update. To further mitigate the risk of infusion related symptoms, the prophylaxis, given before each infusion of BI 836858, was adapted |
| Section to be changed | Section 4.1.4 Drug assignment and administration of doses for each patient |
| Description of change | Text added for clarification: Neutrophils ≥500 /μL (0.5 x 10 <sup>9</sup> /L) and platelets ≥25,000 /μL (25 x 10 <sup>9</sup> /L), unless CTCAE Grade 4 neutropenia or thrombocytopenia was preexistent prior to trial entry. "Patients with active leukemia who go from Grade 3 neutropenia to Grade 4 neutropenia after treatment may continue on study provided there is no evidence of infection or febrile neutropenia. Patients with active leukemia who go from Grade 3 to Grade 4 thrombocytopenia after treatment may continue on study provided that post-transfusion platelet count is at least 20,000/uL before therapy is given." |

BI Trial No.: 1315.1 Doc. No.: c02543230-04 Trial Protocol 

| Number of global amendment | 02 |
|---|---|
| Rationale for change | Clarification |
| Section to be changed | Section 4.1.7 Storage conditions |
| Description of change | Added "- stored in a refrigerator 36-46°F (2-8°C); |
| Description of change | do not freeze". |
| Rationale for change | Clarification |
| Section to be changed | Section 4.2.2.1 Restrictions regarding concomitant |
| Section to be changed | treatment |
| Description of change | The word "the" was removed from text |
| Description of change | The word the was removed from text |
| | Text was modified and added to allow use of |
| | Hydroxyurea as follows: "Prior anti-leukemia |
| | therapy must have been discontinued at least two |
| | weeks before the first administration of the trial |
| | drug (Hydroxyurea may be given <i>during study</i> |
| | participation) until 48 hours before the first |
| | treatment with BI 836858) and the patient must |
| | have recovered from all clinically relevant |
| | reversible toxicities as determined by the |
| | investigator. |
| | investigator. |
| | "For peripheral blood blast control, as this may correlate with the risk of occurrence of infusion related symptoms, hydroxyurea will be allowed (maximum dose of hydroxyurea 3gm daily) before and during study participation. Leukocyte must be ≤ 5,000/µl at start of each administration of BI 836858. During the first two dose cohorts, if in the first cycle more than 2 patients who receive BI 836858 experience a leukocyte count over 40,000/µl indicative of disease progression, then hydroxyurea will be allowed (maximum dose of hydroxyurea 3gm daily) during the week after the first infusion of BI 836858 for all subsequent patients. |
| | If the change of permitting hydroxyurea is implemented and more than 2 of the next 6 patients experience the leukocytosis (40,000/µl indicative of disease progression) and discontinue the due to disease progression in the first cycle, then the eligibility criteria will be modified such that patients requiring hydroxyurea within a week of study entry to maintain WBC <30,000/ul will no longer be eligible. |

BI Trial No.: 1315.1 Doc. No.: c02543230-04 Trial Protocol 

| Number of global amendment | 02 |
|---|---|
| Rationale for change | Clarification and update. To control the WBC, a treatment with hydroxyurea will be allowed. The parallel use of hydroxyurea may allow patients with a proliferative disease to remain on the study. This may also reduce the number of early study withdrawals, especially in the lower dose cohorts, as disease progression may be controlled. |
| Section to be changed | Section 5.1.2.3 Assessment and definition of best overall response |
| Description of change | Language updated for clarification to read as follows: "Response will be assessed according to the criteria from the IWG based on laboratory data from the peripheral blood, bone marrow examination, and clinical examination (at the end of each cycle), e.g. prior to the next dose of BI 836858, at the evaluation for further treatment-visit and, the EOT-visit., and at all follow up visits. Bone marrow examination will be performed before the Cycle 3 and Cycle 5 (5th and 9th administration of BI 836858) (i.e., BM performed on Day 1 (+/-1) of cycles 3 and 5 and treatment started on Day 1 (up to +3) of cycles 3 and 5) and at the discretion of the Investigator, e.g. in case clinical and laboratory examinations of peripheral blood demonstrate that a CR has been achieved, or for assessment of persistent neutropenia, anemia or thrombocytopenia." Treatment Failure: added "Resistant disease: Patient survives ≥7 days post-course of treatment; persistent leukemia in blood or bone marrow. Aplasia: Patient survives ≥7 days post-course of treatment; death while cytopenic, with aplastic bone marrow Indeterminate cause: Patients who die < 7 days posttherapy. Patients who die > 7 days posttherapy with no peripheral blood blasts, but no bone marrow examination. Patients who do not complete the first course of therapy. Morphologic relapse: Reappearance of blasts post-CR in peripheral blood or bone marrow." Progressive Disease: removed "10%" for increase of |

| Number of global amendment | 02 |
|---|---|
| 9 | blast population in bone marrow or peripheral blood |
| | and replaced with "50%". |
| Rationale for change | Clarification and update |
| Section to be changed | |
| Rationale for change | Updated |
| Section to be changed | Section 5.2.2.1 Definitions of adverse events |
| Description of change | Protocol-specified significant events: Updated for patients with impaired liver function at baseline "2.5" was removed and replaced with "5.0" times ULN for AST or ALT is considered a protocol-specified significant event. And "1.5" was removed and replaced with "2.0"ULN for bilirubin protocol-specified significant event. Clarification added that SAEs should be reported "(within 24 hours or the next business day whichever is shorter)". Change of spelling in the word DILI |
| Rationale for change | Clarification and update |
| Section to be changed | Section 5.2.3.1 General safety laboratory parameters |
| Description of change | Text added: "An additional safety lab will be collected on day 2 of Cycle 1 (i.e., 24 hours after the first administration of BI 836858). Other lab tests to be included: haptoglobin, direct Coombs test, bilirubin (direct and indirect) and free hemoglobin. Non pre-existing abnormal laboratory values (CTCAE Grade 3 or higher) will be followed up every 48 hours until these laboratory values are back to at least CTCAE Grade 1." |
| Rationale for change | Update |
| Section to be changed | Section 5.2.5.1 Vital signs |

| Number of global amendment | 02 |
|---|---|
| Description of change | Text was updated: Additional time points for blood pressure and heart rate at the day of administration of BI 836858 are: prior to the start of premedication, prior to the start of BI 836858 infusion, and in 30 ( $\pm 10$ ) minute intervals throughout the course of the and 30 ( $\pm 10$ ), 60 ( $\pm 10$ ), 90 ( $\pm 10$ ), 120 ( $\pm 10$ ), 150 ( $\pm 10$ ) and 180 ( $\pm 10$ ) minutes after start of the infusion of BI 836858 and 60 ( $\pm 10$ ) minutes after the end of the infusion, thereafter every 4-8 hours until at least 24 hours after the start of the infusion. |
| Rationale for change | Clarification and update |
| Section to be changed | Section 5.2.5.2 Physical examination |
| Description of change | Added "height" for clarification of procedures to be performed during a PE. |
| Rationale for change | Clarification |
| Section to be changed | Section 5.3.2.1 Demographics and history |
| Description of change Rationale for change | Updated to include "CRi". Clarification |
| Section to be changed | Section 5.4 Appropriateness of measurements |
| Description of change | References updated removing "R10-4429" and |
| | replacing with "R06-0452". |
| Rationale for change | Update |
| Section to be changed | Section 5.5.1 |

| Number of global amendm | ent | 02 |
|-------------------------|-----|----------------------------------------------|
| | | Operating Procedure (SOP) 001-MCS-36-472_RD- |
| <del></del> | | |
| <del></del> | | |
| <del></del> | | <del></del> |
| | | <del></del> |
| <del></del> | | |
| <u> </u> | | <del></del> |
| | | _ |
| | | <u> </u> |

| Number of global am | endment | 02 |
|-----------------------|---------|-------------------------------------------|
| _ | | |
| - | | |
| _ | | |
| - | | <del></del> |
| - | | |
| - | | |
| _ | | |
| - | | |
| Section to be changed | , | Section 6.2.1 Screening and run-in period |
| Description of change | | Updated to be consistent with Flow Chart: |
| Description of change | , l | "Visit 0" revised to "Visit 1" |
| | | "and baseline conditions" was added to |
| | | Demographics |
| | | Demographics |
| D-4:1- 6 1 | | Clarification |
| Rationale for change | | Clarification |

BI Trial No.: 1315.1 Doc. No.: c02543230-04 Trial Protocol 

| Added Section 6.2.1.1 Rescreening Description of change Added to include rescreening of patients for the trie Section to be change Section 6.2.2.1 Visit 1 and Visit 3 – day of BI 836858 administration (administrations 1-8) Safety lab was updated as follows: "An additional safety lad will be collected on day 2 (i.e., 24 hours after the first administration of BI 836858). Other lab tests to be included: haptoglobin, direct Coombs test, bilirubin (direct and indirect) and free hemoglobin. Non pre-existing abnormal laboratory values (CTCAE Grade 3 or higher) will be followed up every 48 hours until these laboratory values are back to at least CTCAE Grade 1." Physical examination and ECOG text modified for clarification: Physical examination "and ECOG performance score completed" every second cycle beginning with cycle 1Physical exam may be completed up to 2 days prior to administration and ECOG must be completed on the day of the administration.}. Heigh and weight (only at Day 1 of first cycle)—and ECOG performance score. If the first administration is completed within 3 days of the screening visit, these examinations do not need to be repeated. Biomarkers updated with reference to collection time points in Table 3 Clarification and update. The aim is to observe elevated laboratory values earlier and, with additional parameters (e.g. liver enzymes) to better understand the cause of the laboratory values. | Number of global amendment | 02 |
|---|---|---|
| Description of change Added to include rescreening of patients for the trial Rationale for change Update Section to be changed Section 6.2.2.1 Visit 1 and Visit 3 – day of BI 836858 administration (administrations 1-8) | | |
| Rationale for change Section to be changed Section 6.2.2.1 Visit 1 and Visit 3 – day of BI 836858 administration (administrations 1-8) Safety lab was updated as follows: "An additional safety lab will be collected on day 2 (i.e., 24 hours after the first administration of BI 836858). Other lab tests to be included: haptoglobin, direct Coombs test, bilirubin (direct and indirect) and free hemoglobin. Non pre-existing abnormal laboratory values (CTCAE Grade 3 or higher) will be followed up every 48 hours until these laboratory values are back to at least CTCAE Grade 1." Physical examination and ECOG text modified for clarification: Physical examination "and ECOG performance score completed" every second cycle beginning with cycle 1. "Physical exam may be completed up to 2 days prior to administration and ECOG must be completed on the day of the administration." Heigh and weight (only at Day 1 of first cycle). and ECO performance-score. If the first administration is completed within 3 days of the screening visit, these examinations do not need to be repeated. Biomarkers updated with reference to collection time points in Table 3 Clarification and update. The aim is to observe elevated laboratory values earlier and, with additional parameters (e.g. liver enzymes) to better understand the cause of the laboratory values. | | - |
| Section to be changed Section 6.2.2.1 Visit 1 and Visit 3 – day of BI 836858 administration (administrations 1-8) Safety lab was updated as follows: "An additional safety lab will be collected on day 2 (i.e., 24 hours after the first administration of BI 836858). Other lab tests to be included: haptoglobin, direct Coombs test, bilirubin (direct and indirect) and free hemoglobin. Non pre-existing abnormal laboratory values (CTCAE Grade 3 or higher) will be followed up every 48 hours until these laboratory values are back to at least CTCAE Grade 1." Physical examination and ECOG text modified for clarification: Physical examination "and ECOG performance score completed" every second cycle beginning with cycle 1(Physical exam may be completed up to 2 days prior to administration and ECOG must be completed on the day of the administration.), Heigh and weight (only at Day 1 of first cycle). and ECOG performance score. If the first administration is completed within 3 days of the screening visit, these examinations do not need to be repeated. Biomarkers updated with reference to collection time points in Table 3 Clarification and update. The aim is to observe elevated laboratory values earlier and, with additional parameters (e.g. liver enzymes) to better understand the cause of the laboratory values. | | |
| Safety lab was updated as follows: "An additional safety lab will be collected on day 2 (i.e., 24 hours after the first administration of BI 836858). Other lab tests to be included: haptoglobin, direct Coombs test, bilirubin (direct and indirect) and free hemoglobin. Non pre-existing abnormal laboratory values (CTCAE Grade 3 or higher) will be followed up every 48 hours until these laboratory values are back to at least CTCAE Grade 1." Physical examination and ECOG text modified for clarification: Physical examination "and ECOG performance score completed" every second cycle beginning with cycle 1Physical exam may be completed up to 2 days prior to administration and ECOG must be completed on the day of the administration. It fleigl and weight (only at Day 1 of first cycle)and ECOG performance score. If the first administration is completed within 3 days of the screening visit, these examinations do not need to be repeated. Biomarkers updated with reference to collection time points in Table 3 Clarification and update. The aim is to observe elevated laboratory values earlier and, with additional parameters (e.g. liver enzymes) to better understand the cause of the laboratory values. | | |
| Safety lab was updated as follows: "An additional safety lab will be collected on day 2 (i.e., 24 hours after the first administration of BI 836688). Other lab tests to be included: haptoglobin, direct Coombs test, bilirubin (direct and indirect) and free hemoglobin. Non pre-existing abnormal laboratory values (CTCAE Grade 3 or higher) will be followed up every 48 hours until these laboratory values are back to at least CTCAE Grade 1." Physical examination and ECOG text modified for clarification: Physical examination "and ECOG performance score completed" every second cycle beginning with cycle 1. #Physical exam may be completed up to 2 days prior to administration and ECOG must be completed on the day of the administration. Heigh and weight (only at Day 1 of first cycle). *and ECOG performance seere. If the first administration is completed within 3 days of the screening visit, these examinations do not need to be repeated. Biomarkers updated with reference to collection time points in Table 3 Clarification and update. The aim is to observe elevated laboratory values earlier and, with additional parameters (e.g. liver enzymes) to better understand the cause of the laboratory values. | Section to be changed | |
| safety lab will be collected on day 2 (i.e., 24 hours after the first administration of Bl 836858), Other lab tests to be included: haptoglobin, direct Coombs test, bilirubin (direct and indirect) and free hemoglobin. Non pre-existing abnormal laboratory values (CTCAE Grade 3 or higher) will be followed up every 48 hours until these laboratory values are back to at least CTCAE Grade 1." Physical examination and ECOG text modified for clarification: Physical examination "and ECOG performance score completed" every second cycle beginning with cycle 1(Physical exam may be completed up to 2 days prior to administration and ECOG must be completed on the day of the administration.), Heigh and weight (only at Day 1 of first cycle). and ECOG performance score. If the first administration is completed within 3 days of the screening visit, these examinations do not need to be repeated. Biomarkers updated with reference to collection time points in Table 3 Clarification and update. The aim is to observe elevated laboratory values earlier and, with additional parameters (e.g. liver enzymes) to better understand the cause of the laboratory values. | Description of change | |
| clarification: Physical examination "and ECOG performance score completed" every second cycle beginning with cycle 1(Physical exam may be completed up to 2 days prior to administration and ECOG must be completed on the day of the administration.), Height and weight (only at Day 1 of first cycle). and ECOG performance score. If the first administration is completed within 3 days of the screening visit, these examinations do not need to be repeated. Biomarkers updated with reference to collection time points in Table 3 Clarification and update. The aim is to observe elevated laboratory values earlier and, with additional parameters (e.g. liver enzymes) to better understand the cause of the laboratory values. | Description of change | safety lab will be collected on day 2 (i.e., 24 hours after the first administration of BI 836858). Other lab tests to be included: haptoglobin, direct Coombs test, bilirubin (direct and indirect) and free hemoglobin. Non pre-existing abnormal laboratory values (CTCAE Grade 3 or higher) will be followed up every 48 hours until these laboratory values are back to at least CTCAE |
| The aim is to observe elevated laboratory values earlier and, with additional parameters (e.g. liver enzymes) to better understand the cause of the laboratory values. | | clarification: Physical examination "and ECOG performance score completed" every second cycle beginning with cycle 1.—(Physical exam may be completed up to 2 days prior to administration and ECOG must be completed on the day of the administration.)—, Height and weight (only at Day 1 of first cycle).—and ECOG performance score. If the first administration is completed within 3 days of the screening visit, these examinations do not need to be repeated. Biomarkers updated with reference to collection |
| | Rationale for change | Clarification and update. The aim is to observe elevated laboratory values earlier and, with additional parameters (e.g. liver enzymes) to better understand the cause of the |
| <u> </u> | | |
| Section to be changed Section 6.2.3.1 EOT visit | Section to be changed | Section 6.2.3.1 EOT visit |
| <b>Description of change</b> ", PR or CR" deleted | | |
Boehringer Ingelheim
BI Trial No.: 1315.1

| Number of global amendment | 02 |
|---|---|
| Rationale for change | Update |
| Section to be changed | Section 6.2.3.2 Further treatment (Visit 1 and Visit |
| a contract of cont | 2) |
| Description of change | Language updated to: "These visits are only for |
| | those patients with clinical benefit, PR, or CR after |
| | 8 administrations and who are tolerating the |
| | infusions well. Patients can receive further |
| | treatment once the result from the bone marrow |
| | assessment from EOT is available. Procedures |
| | already done at EOT (i.e., safety lab, pregnancy |
| | test) do not need to be repeated at FTE if FTE visit |
| | is within 7 days from EOT." |
| Rationale for change | Clarification and update |
| Section to be changed | Section 6.2.3.3 End of further treatment |
| Description of change | Physical examination language clarification to |
| | include "weight" |
| Rationale for change | Clarification |
| Section to be changed | Section 6.2.3.4 Follow up |
| Description of change | Text added: "Vital status evaluated at each follow |
| | up visit." |
| Rationale for change | Updated |
| Section to be changed | Section 7.3.2.3 Best overall response |
| Description of change | Updated with "or PR" for consistency and |
| | clarification |
| Rationale for change | Clarification |
| Section to be changed | Section 7.3.3 Safety analyses |
| Description of change | MTD determination clarification to be completed |
| | after 2 cycles |
| Rationale for change | Clarification |
| Section to be changed | |
| Rationale for change | Clarification |
| Section to be changed | Section 9.1 Published References |
| Description of change | Reference removed (R10-4429) and added (R01-0787) |
| Rationale for change | Update |
| Section to be changed | Section 10.2 EASTERN COOPERATIVE |
| | ONCOLOGY GROUP (ECOG) Performance |

Boehringer Ingelheim
BI Trial No.: 1315.1

Doc. No.: c02543230-04 Trial Protocol 

| Number of global amendment | 02 |
|----------------------------|---------------------------------------|
| | Status |
| Description of change | Section/Table added for clarification |
| Rationale for change | Clarification |

BI Trial No.: 1315.1 Doc. No.: c02543230-04 Trial Protocol 

| Number of global amendment | 03 |
|---|---|
| Date of CTP revision | 28 April 2016 |
| EudraCT number | N/A |
| BI Trial number | 1315.1 |
| BI Investigational Product(s) | BI 836858 |
| Title of protocol | A Phase I, open label, cohort dose escalation trial |
| Title of protocor | with BI 836858 in patients with refractory or |
| | relapsed acute myeloid leukemia and patients |
| | with acute myeloid leukemia in complete |
| | remission with high risk to relapse |
| | remission with high risk to reliable |
| To be implemented only after | |
| approval of the | |
| IRB/IEC/Competent | |
| Authorities | |
| To be implemented | |
| immediately in order to | |
| eliminate hazard – | |
| IRB / IEC / Competent | |
| Authority to be notified of | |
| change with request for | |
| approval | |
| Can be implemented without | |
| IRB/IEC/ Competent | |
| Authority approval as changes | |
| involve logistical or | |
| administrative aspects only | |
| Section to be changed | Title Page |
| Description of change | Title of trial updated |
| Rationale for change | Updated to include new patient population |
| | "Patients with AML in complete remission (CR) |
| | with high risk to relapse" |
| Section to be changed | Synopsis: title of trial, objectives, No. of patients, |
| | inclusion criteria, test product, duration of |
| | treatment, criteria for efficacy |
| Description of change | Protocol synopsis sections updated to include new |
| | patient population |
| Rationale for change | Revised to include new patient population |
| Section to be changed | Flow Chart |
| Description of change | A new Flow Chart was added for the new patient |
| | population. To differentiate them, now labelled |
| | "Flow Chart A" and "Flow Chart B" plus patient |
| | population. Footnote section in FC - A updated. |
| Rationale for change | Updated to include new patient population |

BI Trial No.: 1315.1 Doc. No.: c02543230-04 Trial Protocol 

| Number of global amendment | 03 |
|---|---|
| Number of global amenument | |
| - | <del> </del> |
| <del></del> | <del></del> |
| Section to be changed | Abbreviations |
| Description of change | Updated with new abbreviations; abbreviation |
| Description of change | definitions revised; abbreviation deleted |
| Rationale for change | Update Update |
| | 1 |
| Section to be changed Description of change | 1.1 Medical Background |
| Description of change | New patient population information added and |
| | differentiated from refractory/relapsed patients. |
| Dationals for shares | Deletion of language to update section. Updated to include new patient population and |
| Rationale for change | medical background information |
| Section to be abanged | |
| Section to be changed Description of change | 1.1 Medical Background Addition of lintuzumab paragraph |
| Rationale for change | To update medical background information |
| Section to be changed | 1.2 Drug Profile |
| i | · |
| Description of change | Investigator brochure reference updated; |
| Dationals for shangs | preliminary data from current study added Updated with new information |
| Rationale for change | 2.1 Rationale for Performing the Trial |
| Section to be changed | <u> </u> |
| Description of change | Section updated and preliminary data added to include new patient population |
| Dationals for shangs | |
| Rationale for change | Updated to support rationale of new patient population |
| Castian to be abanged | 2.1 Rationale for Performing the Trial |
| Section to be changed | Addition of lintuzumab paragraph |
| Description of change | Update Update |
| Rationale for change | 2.2 Trial Objectives |
| Section to be changed | 3 |
| Description of change | Language revised since there will be more than 1 MTD |
| Pationala for change | clarification |
| Rationale for change<br>Section to be changed | 2.3 Benefit – Risk Assessment |
| | Text updated with new patient population; section |
| Description of change | updated/language deleted; new clinical data added |
| Dationals for shangs | Updated to support addition of new patient |
| Rationale for change | population |
| Section to be abanged | |
| Section to be changed | 3.1 Overall Trial Design and Plan Taxt added/deleted and undeted to differentiate |
| Description of change | Text added/deleted and updated to differentiate |
| Dationals for abores | both patient populations Undeted to include new patient population |
| Rationale for change | Updated to include new patient population |

BI Trial No.: 1315.1

| Number of global amendment | 03 |
|---|---|
| Section to be changed | 3.1.1, 4.1.6, 5.2.3.2, 5.2.4, 5.2.5.2, 7.3.2.3, 7.3.6, |
| | and 10.3.2 |
| Description of change | Grammatical and spelling updates |
| Rationale for change | Updates |
| Section to be changed | 3.2 Discussion of Trial Design, Including the |
| | Choice of Control Group |
| Description of change | Text added/deleted and updated to differentiate |
| | both patient populations |
| Rationale for change | Updated to include new patient population |
| Section to be changed | 3.3 Selection of Trial Population |
| <b>Description of change</b> | Text added/deleted to differentiate both patient |
| | populations; number of patients screened and |
| | entered updated |
| Rationale for change | Updated to include new patient population |
| Section to be changed | 3.3.1 Main Diagnosis for Study Entry |
| Description of change | Text added to differentiate both patient |
| | populations; text deleted |
| Rationale for change | Updated to include new patient population |
| Section to be changed | 3.3.2 Inclusion criteria |
| Description of change | Text added to differentiate both patient |
| | populations |
| Rationale for change | Updated to include new patient population |
| Section to be changed | 3.3.3 Exclusion criteria |
| Description of change | Text added/deleted and updated in exclusions # 1, |
| | # 2, # 3, and # 5 to differentiate both patient |
| | populations |
| Rationale for change | Updated to include new patient population |
| Section to be changed | 3.3.3 Exclusion criteria |
| Description of change | Text updated in exclusions # 4 and #19 for |
| | clarification |
| Rationale for change | Clarification and update |
| Section to be changed | 3.3.4.1 Removal of individual patients |
| Description of change | Text added/updated to differentiate expectations |
| | in both patient populations |
| Rationale for change | Updated to include new patient population |
| Section to be changed | 3.3.4.1 Removal of individual patients |
| Description of change | Vital status collection added for clarification |
| Rationale for change | Clarification |
| Section to be changed | 4.1.1 Identity of BI investigational product and |
| | comparator product |
| Description of change | Text added to clarify days when drug |
| | administered |
| Rationale for change | Updated as per new patient population |

**BI Trial No.: 1315.1** 

| Number of global amendment | 03 |
|---|---|
| Section to be changed | 4.1.3 Selection of doses in the trial |
| Description of change | Text added/deleted to differentiate both patient |
| Description of change | populations; new IB reference # included |
| Rationale for change | Text added/deleted to differentiate both patient |
| The country of the co | populations |
| Section to be changed | 4.1.4 Drug assignment and administration of |
| section to be changed | doses for each patient |
| Description of change | Text added/deleted to differentiate both patient |
| bescription of entinge | populations; text updated in premedication and |
| | retreatment sections; text added regarding intra- |
| | patient dose escalation |
| Rationale for change | Updated to include new patient population and to |
| Tanvonare for enange | allow intra-patient dose escalation |
| Section to be changed | 4.1.5.1 Blinding |
| Description of change | Text added to differentiate both patient |
| | populations |
| Rationale for change | Updated to include new patient population |
| Section to be changed | 4.1.8 Drug accountability |
| Description of change | Drug substance added to text for clarification |
| Rationale for change | Updated for clarification |
| Section to be changed | 4.2.1 Rescue medication, emergency procedures, |
| | and additional treatments |
| Description of change | Text deleted for clarification |
| Rationale for change | Updated for clarification |
| Section to be changed | 4.2.2.1 Restrictions regarding concomitant |
| | treatment |
| Description of change | Text updated for clarification |
| Rationale for change | Clarification |
| Section to be changed | 5.1.1 Endpoints of efficacy |
| Description of change | Endpoints modified to differentiate between |
| | patient populations; endpoints deleted; secondary |
| | endpoints changed to further endpoints. |
| | Deleted supportive care endpoint and change |
| | secondary endpoints to further endpoints |
| Rationale for change | Updated to differentiate both patient populations |
| | and to clarify study intended endpoints |
| Section to be changed | 5.1.1 Endpoints of efficacy |
| Description of change | Language on supportive care requirements was |
| D.C. L.C. L | deleted to update endpoints |
| Rationale for change | update |
| | <del></del> |

BI Trial No.: 1315.1 Doc. No.: c02543230-04 Trial Protocol 

| Number of global amendment | 03 |
|---|---|
| g | |
| Section to be changed | 5.1.2.3 Assessment and definition of best overall |
| | response |
| Description of change | Text added for clarification and differentiation of |
| | patient populations; addition of stable disease and |
| | morphologic relapse as it was previously omitted |
| | in error |
| Rationale for change | Updated to differentiate both patient populations |
| | and for further clarification |
| Section to be changed | 5.1.2.3 Assessment and definition of best overall |
| | response |
| Description of change | Language on Stable Disease added for update |
| Rationale for change | Update |
| Section to be changed | 5.1.2.4 Progression free survival (PFS) |
| Description of change | Text added to clarify date of progression/relapse for clarification |
| Rationale for change | Updated for clarification |
| Section to be changed | 5.1.2.5 Time to treatment failure (TTF) |
| Description of change | Text added/deleted to clarify date of |
| Detionals for shares | progression/relapse |
| Rationale for change | Updated for clarification |
| Section to be changed | |
| <del>- +</del> | |
| <del></del> | |
| Description of change | Text added for clarification |
| Rationale for change | Updated to clarify date of progression/relapse |
| Section to be changed | 5.1.2.8 Supportive care requirements |
| Description of change | Section deleted |
| Rationale for change | Deleted as "supportive care requirements" is no |
| v | longer an endpoint |
| Section to be changed | 5.1.2.9 ECOG Performance status |
| Description of change | Section # changed from 5.1.2.9 to 5.1.2.8 |
| Rationale for change | Revised as per deletion of the "supportive care |
| | requirements" |
| Section to be changed | 5.2.1 Endpoints of safety |
| Description of change | Text added/deleted to specify primary and further |
| | safety endpoints |

BI Trial No.: 1315.1 Doc. No.: c02543230-04 Trial Protocol 

| Number of global amendment | 03 |
|---|---|
| Rationale for change | Updated for clarification |
| Section to be changed | |
| Description of change | 5.2.1.1 Dose Limiting Toxicity (DLT) Section subtitle updated with refractory/relapsed |
| Description of change | patient population; Text added/deleted for |
| | clarification |
| D. C. J. C. J. | |
| Rationale for change | Updated to reflect text relevant to refractory/ |
| | relapsed patients |
| Section to be changed | 5.2.1.2 Dose Limiting Toxicity (DLT) for AML |
| | patients in CR |
| Description of change | Section added for inclusion of this patient |
| | population; text added/deleted for clarification |
| | and differentiation of each patient population |
| Rationale for change | Updated to include new patient population |
| Section to be changed | Section 5.2.2 Assessment of adverse events, |
| | 5.2.2.1, 5.2.2.2 |
| Description of change | Sections updated as per new protocol template |
| Rationale for change | Update |
| Section to be changed | 5.2.3.1 General safety laboratory parameters |
| Description of change | Text updated to reflect the new flow chart and |
| | change or clarification in lab test |
| Rationale for change | Clarification |
| Section to be changed | 5.3.2.1 Demographics and history |
| Description of change | Text added/deleted to differentiate patient |
| | population |
| Rationale for change | Updated |
| | _ |
| <del></del> | _ |
| <del> </del> | <del> </del> |
| <del> </del> | <del> </del> |
| <del> </del> | <del> </del> |
| <del></del> | |
| <del></del> | |
| <del></del> | <del></del> |
| | <del></del> |
| <u> </u> | <del>_</del> |


© 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies. All rights reserved.

BI Trial No.: 1315.1 Doc. No.: c02543230-04 Trial Protocol 

| Number of global amendment | 03 |
|---|---|
| 1 tumber of global amenument | |
| <del> </del> | <del></del> |
| <del></del> | <del>- </del> |
| <del></del> | |
| Section to be changed | 6. Investigational Plan sections (6.1, 6.2, 6.2.1, |
| Section to be changed | 6.2.2, 6.2.2.1, 6.2.2.2, 6.2.3 subtitle, 6.2.3.1, |
| | 6.2.3.2, 6.2.4, 6.2.4.1, 6.2.4.2, 6.2.4.3, 6.2.4.4, |
| | 6.2.4.5, 6.2.5 (former 6.2.3.4) and 6.2.6 (former |
| | 6.2.3.5) |
| Description of change | Text in these sections were added/updated to |
| Description of change | differentiate procedures to be performed with |
| | each patient population and to reflect new flow |
| | chart and tables |
| Rationale for change | Update and clarification |
| Section to be changed | 7.1 statistical Design - Model |
| Description of change | Text added to differentiate both patient |
| Description of change | populations |
| Rationale for change | Update |
| Section to be changed | 7.3 Planned Analyses |
| Description of change | Text updated for clarification |
| Rationale for change | Update |
| Section to be changed | 7.3.1 & 7.3.2 Primary and secondary analyses |
| Description of change | Text updated to include both patient populations |
| Rationale for change | Update |
| Section to be changed | 7.3.2.6 Supportive care requirements |
| Description of change | Section deleted |
| Rationale for change | Section deleted as "supportive care requirements" |
| | is no longer an endpoint |
| Section to be changed | 7.3.2.7 ECOG score |
| Description of change | Section # changed from 7.3.2.7 to 7.3.2.6 due to |
| | deletion of previous section |
| Rationale for change | Update |
| Section to be changed | 7.3.3 Safety analyses |
| Description of change | Text updated as per new protocol template |
| | language |
| Rationale for change | Update |
| Section to be changed | 7.3.4 Interim analyses |
| Description of change | Text updated as per new preliminary data |
| | obtained from the refractory /relapsed patient |
| | population |

Boehringer Ingelheim
BI Trial No.: 1315.1

| Number of global amendment | 03 |
|---|---|
| Rationale for change | Update |
| Section to be changed | 7.6 Determination of Sample Size |
| Description of change | Text added and updated to differentiate both |
| | patient populations |
| Rationale for change | Update |
| Section to be changed | 8.4.1 Listedness |
| Description of change | IB reference # updated |
| Rationale for change | Update |
| Section to be changed | 9.1 & 9.2 Published and Unpublished References |
| Description of change | References added:R10-2947, R11-4695, and |
| | c02324887-03 |
| Rationale for change | Update |
| Section to be changed | 10.2 ECOG |
| Description of change | Reference # added for clarification |
| Rationale for change | Update |



### APPROVAL / SIGNATURE PAGE

Document Number: c02543230 Technical Version Number: 1.0

**Document Name:** clinical-trial-protocol-rev3

**Title:** A Phase I, open, cohort dose escalation trial with BI 836858 in patients with refractory or relapsed acute myeloid leukemia

## Signatures (obtained electronically)

| Meaning of Signature | Signed by | Date Signed |
|----------------------------------------|-----------|------------------------|
| Approval–Clinical Monitor | | 28 Apr 2016 22:06 CEST |
| Author-Trial Statistician | | 29 Apr 2016 11:47 CEST |
| Approval-Therapeutic Area | | 29 Apr 2016 14:19 CEST |
| Approval-Translational Medicine Expert | | 29 Apr 2016 14:37 CEST |
| Approval-Team Member Medicine | | 29 Apr 2016 17:02 CEST |

Boehringer IngelheimPage 2 of 2Document Number: c02543230Technical Version Number: 1.0

# (Continued) Signatures (obtained electronically)

| Meaning of Signature S | Signed by | <b>Date Signed</b> |
|------------------------|-----------|--------------------|
|------------------------|-----------|--------------------|